#### The GlaxoSmithKline group of companies

| Division | ŀ | Worldwide Development |
|---|---|---|
| Information Type : Reporting and Analysis Plan (RAP) | | Reporting and Analysis Plan (RAP) |

| Title | : | A Phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with hepatic impairment and matched, healthy control participants with normal hepatic function |
|---|---|---|
| <b>Compound Number</b> | : | GSK1278863 |
| Effective Date | : | 22-NOV-2017 |

#### **Description:**

• The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in Clinical Pharmacology Study Report for Protocol 200231.

#### **Author's Name and Functional Area:**

| PPD | 03-OCT-2017 |
|---------------------------------------------------------|-------------|
| Associate Manager Statistics (Clinical Statistics, GSK) | 03-001-2017 |
| PPD | 03-OCT-2017 |
| Manager, Clinical Pharmacology (GSK) | 03-001-2017 |
| PPD | 03-OCT-2017 |
| Pharmacokineticist (Biostatistics, PPD) | 03-001-2017 |
| PPD | 03-OCT-2017 |
| Biostatistician (Early Development Services, PPD) | 03-001-2017 |

### Approved by:

| PPD | 22-NOV-2017 |
|---|---|
| Director, Statistics & Programming (Clinical Statistics, GSK) | 22-NOV-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### **TABLE OF CONTENTS**

| | | | | | | PAGE |
|---|---|---|---|---|---|---|
| 1. | REPC | RTING & | ANALYSIS | S PLAN SYN | POSIS | 4 |
| 2. | STIMM | MADV OF | KEN DDU. | TOCOL INE | DRMATION | 7 |
| ۷. | 2.1. | | | | d Statistical Analysis Plan | |
| | 2.1. | Study Of | bioctivo(c) | and Endnoir | u Statisticai Ariaiysis Fiari | |
| | 2.2. | Study D | ojective(s)<br>seign | and Endpoi | nt(s) | Ω<br>Ω |
| | 2.4. | | | | | |
| 3. | | | | | | |
| | 3.1. | | | | | |
| | 3.2. | Final An | alyses | | | 11 |
| 4. | ANAL | YSIS POF | PULATION | S | | 12 |
| | 4.1. | Protocol | Deviations | 3 | | 13 |
| 5. | CONS | SIDERATION | ONS FOR | DATA ANAI | YSES AND DATA HANDLING | |
| 0. | | | | | | 14 |
| 6. | CTUD | V DODLII | ATIONI AN | IALVECE | | 15 |
| Ο. | 6.1. | | | | | |
| | 0.1. | Overviev | V OI PIAIIII | eu Analyses | | 13 |
| 7. | | | | | | |
| | 7.1. | | | | | |
| | 7.2. | | | | | |
| | | 7.2.1. | | | Pharmacokinetic Analyses | |
| | | | 7.2.1.1. | | entration Measures | |
| | | | 7.2.1.2. | | kinetic Parameters | 17 |
| | | | | 7.2.1.2.1. | | |
| | | | | | Parameters | 17 |
| | | | | 7.2.1.2.2. | | 4.0 |
| | | | | | Pharmacokinetic Parameters | |
| | 7.3. | | codynamic | Analyses | | 21 |
| | | 7.3.1. | Overview | of Planned | Pharmacodynamic Analyses | 21 |
| | | | 7.3.1.1. | | dynamic Parameters | 21 |
| | | | | 7.3.1.1.1. | , | |
| | | | | | Parameters | 21 |
| 8. | SAFF | TY ANAI Y | YSES | | | 23 |
| О. | 8.1. | | | | vents Analyses | |
| | 8.2. | | | | aboratory Analyses | |
| | 8.3. | | | | ety Analyses | |
| _ | | | | | | |
| 9. | KEFE | RENCES. | | | | 26 |
| 10. | | | | | | |
| | 10.1 | | | | Management | |
| | 10.2 | | x 2: Time 8 | & Events | | 29 |
| | | 10.2.1 | | | e & Events | |
| | 10.3 | Appendi | x 3: Treatn | nent States | | 32 |


| 2 | n | Λ | 23 | 4 |
|---|---|---|-----|---|
| | U | u | 2.0 | ) |

| | 10.3.1 | Treatment State | es for AE Data | 32 |
|---|---|---|---|---|
| 10.4 | Appendi | 4: Data Display | Standards & Handling Conventions | 33 |
| | 10.4.1 | | nt & Display Descriptors | |
| | 10.4.2 | Baseline Definit | tion & Derivations | 33 |
| | | 10.4.2.1 Base | eline Definitions | 33 |
| | | | vations and Handling of Missing Baseline | |
| | | | a | |
| | 10.4.3 | | ess & Standards | |
| 10.5 | Appendix 5: Derived and Transformed Data | | | |
| | 10.5.1 | | | |
| | 10.5.2 | | on | |
| | 10.5.3 | | | |
| 10.6 | | | Vithdrawals & Handling of Missing Data | |
| | 10.6.1 | | ndrawals | |
| | 10.6.2 | | ssing Data | |
| | | | dling of Missing Dates | |
| | | | dling of Partial Dates | |
| | | | dling of PK Concentration Data | 42 |
| | | | dling of Missing Data for Statistical | |
| | | Anal | lysis | 42 |
| 10.7 | | | otential Clinical Importance | |
| | 10.7.1 | | Jes | |
| | 10.7.2 | | | |
| | 10.7.3 | | | 44 |
| 10.8. | | | king and Diagnostics for Statistical | |
| 10.9. | | | s & Trade Marks | |
| | 10.9.1 | | | |
| | 10.9.2 | | | |
| 10.10 | | | ı Displays | |
| | 10.10.1 | | umbering | |
| | 10.10.2 | | | |
| | 10.10.3 | | on Tables | |
| | 10.10.4 | • | | |
| | 10.10.5 | | ic Tables | |
| | 10.10.6 | | ic Figures | |
| | 10.10.7 | | mic Tables | |
| | 10.10.8 | Pharmacodyna | mic Figures | |
| | 10 10 9 | ICH Listings | | 55 |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe: |
| | <ul> <li>The planned analyses and output to be included in the Clinical<br/>Pharmacology Study Report for Protocol 200231. This RAP is intended to<br/>describe the safety and pharmacokinetic (PK) analyses required for the<br/>study which will be provided to the study team members to convey the<br/>content of the reporting efforts, specifically Statistical Analysis Complete<br/>(SAC).</li> </ul> |
| Protocol | This RAP is based on original protocol (Dated: [23-May-2017]) for study 200231 [GlaxoSmithKline Document Number: 2016N305941_00]. |
| Primary<br>Objectives | To compare plasma PK parameters of daprodustat and its six metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13)) in participants with hepatic impairment to healthy controls matched in gender, age, and body mass index (BMI). |
| | To evaluate the impact of hepatic impairment on the plasma protein binding and unbound concentration of daprodustat in plasma. |
| Primary<br>Endpoints | <ul> <li>Daprodustat and its metabolites in plasma area under the concentration-time curve from time zero (predose) extrapolated to infinite time [AUC (0-∞)], percentage of AUC (0-∞) obtained by extrapolation (%AUCex), time zero (predose) to time of last quantifiable concentration [AUC(0-t)], maximum observed concentration (Cmax) following a single oral dose of daprodustat, apparent terminal phase half-life (t½), and time of occurrence of Cmax (Tmax) following a single oral dose of daprodustat.</li> </ul> |
| | <ul> <li>Unbound concentration and unbound fraction in plasma of daprodustat at 3,<br/>12, and 24 hours (h) post dose (as data permit).</li> </ul> |
| Secondary<br>Objectives | To characterize the effect of hepatic impairment on the pharmacodynamics (PD) effect of daprodustat. |
| | To assess the safety and tolerability of a single 6 mg dose of daprodustat. |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Secondary<br>Endpoints | <ul> <li>Maximum observed erythropoietin concentration (Cmax, EPO), Time of the<br/>maximum observed erythropoietin concentration (Tmax, EPO) and<br/>erythropoietin area under the concentration-time curve from time zero (pre-<br/>dose) to the last time of quantifiable erythropoietin concentration [AUC (0-t,<br/>EPO)].</li> </ul> |
| | Safety and tolerability parameters, including adverse events and clinical laboratory tests. |
| Study Design | <ul> <li>A phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with moderate (Part 1) and either mild or severe (Part 2) hepatic impairment and matched, healthy control participants with normal hepatic function.</li> <li>Part 1:</li> </ul> |
| | <ul> <li>Part 1 will include 2 cohorts. Cohort 1 includes participants with moderate<br/>hepatic impairment, and Cohort 2 includes matched healthy control<br/>participants.</li> </ul> |
| | <ul> <li>Healthy control participants (n=8) will be matched in gender, age (±10 years), and BMI (±15%) to participants with moderate hepatic impairment (n=8; Child-Pugh score of 7-9).</li> </ul> |
| | All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state. |
| | Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 1 of the study. |
| | Part 2: |
| | <ul> <li>Part 2 will include 2 cohorts. Cohort 3 includes participants with either mild<br/>or severe hepatic impairment, and Cohort 4 includes matched healthy<br/>control participants.</li> </ul> |
| | <ul> <li>Healthy control participants (n=8) will be matched in gender, age (±10 years), and BMI (±15%) to participants with either mild impairment (Child-Pugh score of 5-6) or participants with severe impairment (Child-Pugh score of 10-13) (n=8).</li> </ul> |
| | All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state. |
| | Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 2 of the study. |
| | All participants' total involvement with the study will be up to 7 weeks. |
| Planned<br>Analyses | <ul> <li>An informal interim analysis of the primary PK endpoints of AUC (0-∞),<br/>AUC(0-t) and Cmax will be conducted for completion of Part 1 of the study.</li> </ul> |
| , | The final planned analyses will be performed, as defined in this RAP document, after database freeze has been declared. |
| | Safety and PK/PD data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data |

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| | Standards Library (IDSL) standards. |
| Analysis<br>Population | Screened Population: All participants who were screened will be considered for this population. This population will be used for summarizing screening status. |
| | Enrolled Population: All participants who were successfully screened and enrolled for the trial and for whom a record exists on the study database. This population will be used for summarize number of subjects by Country and Site ID and age ranges. |
| | Safety Population: All participants who received at least 1 dose of study medication. This will be the primary population for the safety analyses. |
| | PK Population: All participants in the 'Safety Population' for whom a PK sample has been obtained and analyzed will be included in the PK population. This population will be used in the evaluation of PK data. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PK data. |
| | PD Population: All participants in the 'Safety Population' who had at least 1 PD assessment. PD samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PD data. |
| Hypothesis | No formal hypotheses will be tested. |
| Interim<br>Analyses | An informal interim analysis of the primary PK endpoints AUC $(0-\infty)$ , AUC $(0-t)$ and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria: |
| | ➢ If a < 2-fold change in daprodustat exposure (AUC) is observed in<br>participants with moderate hepatic impairment compared to the<br>healthy matched control group, the study may enrol participants<br>with severe hepatic impairment and a healthy, matched control<br>group. |
| | ▶ If a ≥ 2-fold change in daprodustat exposure (AUC) is observed<br>in participants with moderate hepatic impairment compared to the<br>healthy matched control group, the study may enrol participants<br>with mild hepatic impairment and a healthy, matched control group. |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The parameters "Emax" and "AUC (E, last)" in the list of secondary endpoints in the protocol have been replaced/added with "Cmax, EPO", "Tmax, EPO" and "AUC (0-t, EPO)", respectively. These new parameters provide a more accurate reflection of the scope for the PD analysis. There were no other changes or deviations to the originally planned statistical analysis specified in the protocol [Dated: 23-May-2017].

## 2.2. Study Objective(s) and Endpoint(s)

| Obj | jectives | Endpoints |
|---|---|---|
| Pri | mary Objectives | Primary Endpoints |
| | To compare plasma PK parameters of daprodustat and its six metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13)) in participants with hepatic impairment to healthy controls matched in gender, age, and body mass index (BMI). | plasma area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC (0-∞)], percentage of AUC(0-∞) obtained by extrapolation (%AUCex), time zero (pre-dose) to last time |
| • | To evaluate the impact of hepatic impairment on the plasma protein binding and unbound concentration of daprodustat in plasma. | <ul> <li>Unbound concentration and unbound fraction<br/>in plasma of daprodustat at 3, 12 and 24 h<br/>post dose (as data permit).</li> </ul> |
| Sec | condary Objectives | Secondary Endpoints |
| • | To characterize the effect of hepatic impairment on the PD effect of daprodustat. | <ul> <li>Maximum observed erythropoietin<br/>concentration (Cmax, EPO), Time of the<br/>maximum observed erythropoietin<br/>concentration (Tmax, EPO) and<br/>erythropoietin area under the concentration-<br/>time curve from time zero (pre-dose) to the<br/>last time of quantifiable concentration [AUC<br/>(0-t, EPO)].</li> </ul> |
| • | To assess the safety and tolerability of a single 6 mg dose of daprodustat. | <ul> <li>Safety and tolerability parameters, including<br/>adverse events and clinical laboratory tests.</li> </ul> |

## 2.3. Study Design

| Overview of Study Design and Key Features | |
|---|---|
| Design Features | A phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with moderate (Part 1) and either mild or severe (Part 2) hepatic impairment and matched, healthy control participants with normal hepatic function. |

#### **Overview of Study Design and Key Features**

#### Part 1:

Part 1 will include 2 cohorts. Cohort 1 includes participants with moderate hepatic impairment, and Cohort 2 includes matched healthy control participants.

Healthy control participants (n=8) will be matched in gender, age  $(\pm 10 \text{ years})$ , and BMI  $(\pm 15\%)$  to participants with moderate hepatic impairment (n=8; Child-Pugh score of 7-9).

All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state.

Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 1 of the study.

#### Part 2:

Part 2 will include 2 cohorts. Cohort 3 includes participants with either mild or severe hepatic impairment, and Cohort 4 includes matched healthy control participants.

Healthy control participants (n=8) will be matched in gender, age ( $\pm 10$  years), and BMI ( $\pm 15\%$ ) to participants with either mild impairment (Child-Pugh score of 5-6) or participants with severe impairment (Child-Pugh score of 10-13) (n=8).

All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state.

Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 2 of the study.

All participant's total involvement with the study will be up to 7 weeks.

#### Dosing

#### Part 1

All participants will be administered 6 mg of daprodustat as a single oral dose, with assessments conducted for up to 48 h post dosing (Please refer to Appendix 2)

#### Part 2

If conducted, all participants will be administered 6 mg of daprodustat as a single oral dose, with assessments conducted for up to 48 h post dosing.

## Treatment Assignment

 Part 1 consists of up to 16 participants (8 in each cohort, excluding possible replacements).

| Overview of Study Design and Key Features | |
|---|---|
| | <ul> <li>Part 2 consists of up to 16 participants (8 in each cohort, excluding possible replacements).</li> <li>All participants will receive the same treatment of a single oral 6 mg dose of daprodustat.</li> </ul> |
| Interim Analyses | <ul> <li>An informal interim analysis of the primary PK endpoints AUC (0-∞), AUC(0-t) and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria:</li> <li> If a &lt; 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with severe hepatic impairment and a healthy, matched control group. </li> <li> If a ≥ 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with mild hepatic impairment and a healthy, matched control group. </li> </ul> |

## 2.4. Statistical Hypotheses

No formal hypotheses will be tested for this study. An estimation approach will be used to evaluate the effect of hepatic impairment (i.e., moderate and potentially either mild or severe) on the PK of daprodustat. The primary comparisons of interest are the single dose PK parameters, including Cmax and AUC of daprodustat in each hepatic impaired cohort compared to the normal hepatic function cohort.

The point estimates of the geometric least squares (GLS) mean ratio for the PK parameters and associated 90% confidence intervals (CIs) will be provided for cohort comparisons (hepatically impaired: healthy participants). The PK parameters will be log-transformed prior to analysis and cohort comparisons will be expressed as ratios on the original scale. %AUCex and Tmax and will be summarized descriptively.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

An informal interim analysis of the primary endpoints AUC  $(0-\infty)$ , AUC(0-t) and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria:

- If a < 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with severe hepatic impairment and a healthy, matched control group.
- If a ≥ 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with mild hepatic impairment and a healthy, matched control group.

#### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Screened Population | All participants who were screened will be considered for this population. This population will be used for summarizing screening status. | Screen Failure |
| Enrolled Population | All participants who were successfully screened and enrolled for the trial and for whom a record exists on the study database. This population will be used for summarize number of subjects by Country and Site ID and age ranges. | Study Population |
| Safety Population | All participants who received at least one dose of study medication. This will be the primary population for the safety analyses. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK Population | All participants in the 'Safety Population' for whom a PK sample has been obtained and analyzed will be included in the PK population. This population will be used in the evaluation of PK data. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PK data. | • PK |
| PD Population | All participants in the 'Safety Population' who had at least 1 PD assessment. PD samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PD data. | • PD |

#### NOTES:

• Please refer to Appendix 10 which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarized and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
  - o This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

### Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Treatment States and Phases |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |

#### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Analyses

The study population displays will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population displays, with full details of data displays being presented in Appendix 10: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Displa | ys Generated |
|---|---|---|
| | Table | Listing |
| Subject Disposition | | |
| Subject Disposition | Y | |
| Reasons for Screening Failures [1] | Υ | Υ |
| Reasons for Withdrawals | | Υ |
| Important Protocol Deviations | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | | Υ |
| Demography | | |
| Demographic Characteristics | Y | Υ |
| Race & Racial Combinations | Y | Υ |
| Study Populations | Υ | Υ |
| Summary of Number of Subjects by Country and Site ID | Y | |
| Summary of Age Ranges | Y | |
| Summary of Child-Pugh score | Υ | Υ |
| Medical/Surgical History & Concomitant Medications | | |
| Medical/Surgical History | | Υ |
| Concomitant Medication | Y | Y |
| Exposure and Treatment Compliance | | |
| Exposure to Study Treatment | | Υ |

#### NOTES:

<sup>•</sup> Y = Yes display generated.

<sup>[1]</sup> Conditional displays, if data is available table and listing will be generated.

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Interim Analyses

An informal interim analysis of the primary PK endpoints AUC (0-∞), AUC(0-t) and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria:

- If a < 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with severe hepatic impairment and a healthy, matched control group.
- If a ≥ 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with mild hepatic impairment and a healthy, matched control group.

### 7.2. Pharmacokinetic Analyses

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of Clinical Pharmacology Sciences and Study Operations (CPSSO), GlaxoSmithKline.

The merge of PK concentration data and CRF data will be performed by PPD Programming under the direct auspices of Clinical Programming, GlaxoSmithKline.

Derivation of PK parameters will be performed by PPD PK group under the direct auspices of Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

Statistical analysis of PK data and parameters will be performed by PPD Statistics and Programming under the direct auspices of Clinical Statistics, GlaxoSmithKline.

#### 7.2.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK population, unless otherwise specified.

Table 3 provides an overview of the planned non-compartmental PK analyses of daprodustat and its six metabolites, (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6) and GSK2531401 (M13)) with full details being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Display Type | | | U | Intran | sforme | ed | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | | Summary | | Individual | | Stats | | Summary | | Individual | | | |
| | Analysis | | | | Analysis | | | | | | | | | |
| | Т | F | L | Т | F | F | L | T | F | L | T | F | F | Г |
| PK Concentrations | | | | <b>Y</b> [3] | <b>Y</b> [1]<br>[2] | <b>Y</b> [1] | <b>Y</b> [3] | | | | | | | |
| Plasma PK<br>Parameters | <b>Y</b> [4] | | | Υ | | | Υ | <b>Y</b> [4] | | Υ | Y | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Logarithmic plots will be created on the same display.
- [2] Separate mean and median plots will be generated.
- [3] Unbound PK Concentrations for Daprodustat only will be summarized on a separate display.
- [4] Supportive SAS Output from Statistical Analysis.

#### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3. Reporting Process & Standards).

#### 7.2.1.2. Pharmacokinetic Parameters

#### 7.2.1.2.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3. Reporting Process & Standards).
- Plasma concentration-time data for daprodustat and its six predominant metabolites will be analysed by non-compartmental methods according to current working practices with WinNonlin 6.4 or higher.
- Non-compartmental analysis will be performed in accordance with GSK PK Guidance document GUI\_51487.
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.
- PK parameters described in Table 4 will be determined from plasma concentration-time data as data permits.

 Table 4
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid (daprodustat and its six metabolites). |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity calculated as: |
| | AUC(0-∞) = AUC(0-t) + C(t) / lambda_z<br>(daprodustat and its six metabolites) |
| | where C(t) is the last measurable concentration. |
| %AUCex | The percentage of AUC $(0-\infty)$ obtained by extrapolation (%AUCex) will be calculated as: |
| | [AUC (0-∞) – AUC(0-t)] / AUC (0-∞) x 100 |
| | (daprodustat and its six metabolites) |
| Cmax | Maximum observed plasma concentration, determined directly from the concentration-time data. (daprodustat and its six metabolites) |
| Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. (daprodustat and its six metabolites) |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. (daprodustat and its six metabolites) |
| t½ | Apparent terminal phase half-life will be calculated as: |
| | t½ = In2 / Lambda_z |
| | (daprodustat and its six metabolites) |
| fu | Unbound fraction (fu) of daprodustat will be calculated using the total and unbound plasma concentration of daprodustat generated at 3, 12 and 24 h post dose for both normal and hepatic impaired participants using the following formula: |
| | Fu=Cunbound/Ctotal |
| free AUC(0-t) | AUC(0-t) * fu (daprodustat) |

| Parameter | Parameter Description |
|---------------|-----------------------------|
| free AUC(0-∞) | AUC(0-∞) * fu (daprodustat) |
| free Cmax | Cmax * fu (daprodustat) |

#### 7.2.1.2.2. Statistical Analysis of Pharmacokinetic Parameters

For each of the parameters AUC (AUC( $0-\infty$ ), AUC (0-t) and %AUCex)-total and free, t½, Tmax and Cmax-total and free the following summary statistics will be calculated and tabulated by each cohort:

- Untransformed Data: N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum and maximum.
- **Log**<sub>e</sub>-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of log<sub>e</sub>-transformed data and between subject geometric coefficient of variation (%CVb).

The following PK statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles). Pharmacokinetic analysis and Statistical analyses of the PK parameter data will be the responsibility of PPD.

#### **Planned Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

Plasma primary PK endpoints include AUC (0-t), AUC (0-∞), Cmax and t½, as data permit

#### **Model Specification**

• The log-transformed AUC(0-t), AUC (0-∞), Cmax and t½ values for daprodustat and metabolites will be analyzed separately using analysis of variance (ANOVA) as appropriate to the study design, fitting a fixed effect term for cohort. Point estimates and 90% CIs for the differences of interest (hepatically impaired versus healthy participants) will be constructed using the residual variance.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios for the hepatically impaired versus healthy participants and 90% CI for the ratios of AUC (0-t), AUC (0-∞). Cmax and t½ for daprodustat and metabolites.

#### Endpoint(s)

Tmax

#### **Planned Pharmacokinetic Statistical Analyses**

#### **Model Specification**

• If data permit, Tmax will be analyzed nonparametrically using the Mann Whitney U test (Wilcoxon rank sum test). The point estimates and 90% CI for the median differences will be derived for hepatic impairment and healthy participants based on Hodges-Lehmann estimation.

#### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• The point estimates and 90% confidence intervals for the median differences will be calculated for the cohort difference (hepatically impaired – healthy participants).

#### **Sensitivity Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

• AUC(0-t), AUC(0-∞), Cmax and t1/2

#### **Model Specification**

 The log-transformed AUC(0-t), AUC(0-∞), Cmax and t½ values for daprodustat and metabolites will be analyzed separately using analysis of covariance (ANCOVA) as appropriate to the study design, fitting fixed effect terms for cohort, gender, age and BMI. Point estimates and 90% CIs for the differences of interest (hepatically impaired versus healthy participants) will be constructed using the residual variance.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Statistical analysis by ANCOVA will be presented in tabular format with geometric mean ratios for the difference between participants with hepatically impairment and healthy participants, and 90% CI for the ratios of AUC(0-t), AUC(0-∞), Cmax and t½ for daprodustat and metabolites.

#### 7.3. Pharmacodynamic Analyses

#### 7.3.1. Overview of Planned Pharmacodynamic Analyses

The PD analyses will be based on the PD population, unless otherwise specified.

Table 5 provides an overview of the planned PD analyses, with full details being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Pharmacodynamic Analyses

| Display Type | Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Absolute Change from Baseline | | | | | | | | | | | | | |
| | Stat | Stats Analysis Summary Individual | | | | | | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | T | F | F | L | Т | F | L | T | F | F | L |
| PD Concentrations | | | | Υ | <b>Y</b> [1][2] | <b>Y</b> [1] | Υ | | | | | | | |
| PD Parameters | | | · | Υ | Y | | Y | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.3.1.1. Pharmacodynamic Parameters

#### 7.3.1.1.1. Deriving Pharmacodynamic Parameters

- Although erythropoietin (EPO) is an endogenous substance, the plasma concentrations of erythropoietin will not be corrected for baseline endogenous levels Pharmacodynamic analysis will be performed on uncorrected (absolute erythropoietin concentrations) data only.
- Maximum observed erythropoietin concentration (Cmax, EPO), Time of the
  maximum observed erythropoietin concentration (Tmax, EPO) and area under the
  concentration-time curve from time zero (pre-dose) to the last time of quantifiable
  erythropoietin concentration [AUC (0-t, EPO)] will be listed and summarised if
  data is available.
- Pharmacodynamic parameters described in Table 6 will be determined from plasma absolute erythropoietin concentration-time data as data permits.

Linear and Semi-Logarithmic plots will be created on the same display.

<sup>[2]</sup> Separate mean and median plots will be generated.

## Table 6 Derived Pharmacodynamic Parameters

| Parameter | Parameter Description |
|---|---|
| Cmax, EPO | Maximum observed EPO concentration |
| Tmax, EPO | Time of the maximum observed EPO concentration |
| AUC (0-t, EPO) | Area under the concentration-time curve from time zero (pre-dose) to the last time of quantifiable erythropoietin concentration |

#### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

#### 8.1. Overview of Planned Adverse Events Analyses

Adverse Events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary and summarized by cohort.

Counting of AEs will be based on the number of subjects – not the number of AEs. For example, if a subject experiences the same AE (i.e. same preferred term) more than once, they are counted only once under the count for the preferred term. If a subject experiences more than one AE in a particular system organ class (SOC), they will only be included once in the count for the SOC, but will appear in the count for each appropriate preferred term within the SOC. Therefore, the sum of the numbers of subjects with each preferred term event within a SOC may exceed the total number of subjects with at least one event.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 7 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | Absolute | | |
|---|---|---|---|
| | Sun | nmary | Individual |
| | T | F | L |
| Adverse Events (AEs) | | | |
| All AEs | Υ | | Υ |
| Serious AEs | Υ | | Υ |
| Drug Related AEs | Υ | | Y |
| AEs leading to withdrawal | Υ | | Y |
| Summary of Common (>=25%) Non-serious Adverse Events by System Organ Class and Preferred Term | Υ | | |
| Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Υ | | |
| Relationship Between System Organ Class and Verbatim Text | | | Y |
| Subject Numbers for Individual Adverse Events | | | Y |
| AEs of special interest [1] | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Conditional displays, if data is available listing will be generated.

#### 8.2. Overview of Planned Clinical Laboratory Analyses

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 8 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| Display Type | Sur | mmary | Individual | Sun | nmary | Individual |
| | Т | F | L | T F | | L |
| Chemistry | | | | | | |
| Clinical Chemistry | Υ | | Υ | Υ | | |
| Clinical Chemistry (Values Outside the PCI Range) | | | Y | | | |
| Haematology | | | | | | |
| Haematology | Υ | | Y | Υ | | |
| Haematology (Values Outside the PCI Range) | | | Y | | | |
| Urinalysis | | | | | | |
| Urinalysis | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 8.3. Overview of Planned Other Safety Analyses

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays

Table 9 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ | | Abso | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| Display Type | Sur | nmary | Individual | Summary | | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Y | | | |
| ECG Values | Υ | | Y | Υ | | |
| ECG Values Outside the PCI Range | | | Y | | | |
| Maximum QTc Values Post-Baseline Relative to Baseline by Category | | | | Υ | | |
| Maximum Increase in QTc Values Post-<br>Baseline Relative to Baseline by | | | | Υ | | |


200231

| Endpoint / Parameter/ | | Abso | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| Display Type | Sui | mmary | Individual | Sum | mary | Individual |
| | Т | F | L | Т | F | L |
| Category | | | | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | |
| Vital Signs Measurements Outside the PCI Range | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9. REFERENCES

GlaxoSmithKline Document Number 2016N305941\_00 (Original – 23-MAY-2017): A Phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with hepatic impairment and matched, healthy control participants with normal hepatic function.

GUI 137354, Information for Authors: Reporting and Analysis Plan (RAP), Global

GUI 51487, Non-Compartmental Analysis of Pharmacokinetic Data, CPMS Global

SOP\_54838, Development, Review & Approval of Reporting & Analysis Plan (RAP), Global

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4: A | Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5: | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General |
| | Study Population |
| | Safety |
| | Pharmacokinetic |
| | Pharmacodynamic |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| | <ul> <li>Handling of Missing Dates</li> </ul> |
| | <ul> <li>Handling of Partial Dates</li> </ul> |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP Appe | endices |
| Section 10.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 10.10 | Appendix 10: List of Data Displays |

## 10.1 Appendix 1: Protocol Deviation Management

There are no pre-defined categories leading to exclusion from the PK population but all protocol deviations will be reviewed on a case-by-case basis.

No subjects will be excluded from the safety population.

## 10.2 Appendix 2: Time & Events

#### 10.2.1 Protocol Defined Time & Events

| Procedure | Screening <sup>1</sup> | Day -1 | Pre-Dose | 0 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 36 h | 48 h | Follow-up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | Х | | | | | | | | | | | | | | | | | |
| Inclusion & Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | | |
| Demography | Χ | | | | | | | | | | | | | | | | | |
| Full physical exam | Χ | | | | | | | | | | | | | | | | | |
| Medical<br>history | Χ | | | | | | | | | | | | | | | | | |
| Past/current medications | Χ | | | | | | | | | | | | | | | | | |
| Laboratory assessments 3 | X | | | | | | | | | | | | | | | | Χ | Х |
| Drug/Alcohol<br>Screen | Х | Х | | | | | | | | | | | | | | | | |
| 12-lead ECG | Χ | Χ | | | | | | | | | | | | | | | Χ | Х |
| Vital Signs<br>and Weight | Χ | Х | | | | | | | | | | | | | | | Х | Х |
| Pregnancy<br>Test | X <sup>4</sup> | X <sup>4</sup> | | | | | | | | | | | | | | | | |

| Procedure | Screening <sup>1</sup> | Day -1 | Pre-Dose | 0 h | 0.5 h | 4 <b>t</b> | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 36 h | 48 h | Follow-up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Females<br>only:<br>Estrogen and<br>FSH <sup>5</sup> | Х | | | | | | | | | | | | | | | | | |
| Admission to Unit | | Х | | | | | | | | | | | | | | | | |
| Brief Physical<br>Exam | | Х | | | | | | | | | | | | | | | Χ | Х |
| Administratio n of daprodustat | | | | Х | | | | | | | | | | | | | | |
| PK blood sampling | | | Х | | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | |
| Protein binding sample | | | Х | | | | | | Х | | | | | Х | Х | | | |
| EPO blood sampling | | | Х | | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | |
| Adverse<br>Events<br>Assessment | Χ | X | Х | Х | X | X | Χ | X | Χ | Χ | Х | X | X | Χ | Х | Х | Х | X |
| Review<br>Concomitant<br>Medications | | X | X | | | | | | | | | | | | Х | | X | X |
| Discharge from Unit | | | | | | | | | | | | | | | | | Χ | |


200231

<sup>&</sup>lt;sup>1</sup> All participants will undergo screening assessments within 28 days of enrolment.

<sup>&</sup>lt;sup>2</sup> A follow-up visit will occur 10-14 days after the dose of study treatment.

<sup>&</sup>lt;sup>3</sup> Laboratory assessment guidance can be found in Protocol Appendix 3.

<sup>&</sup>lt;sup>4</sup> For women of childbearing potential that are not using an approved method of contraception (see Protocol Appendix 6), one negative pregnancy test between Day -7 and Day -4 AND another negative pregnancy test on Day -1 is required. Additional guidance can be found in Protocol Section.9.5.5.

<sup>&</sup>lt;sup>5</sup> All females are to have estrogen and FSH measured at screening.

## 10.3 Appendix 3: Treatment States

#### 10.3.1 Treatment States for AE Data

Assessments and events will be classified according to date of occurrence relative to the start and/or stop date of the study treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before the treatment stop date 2 days |
| | Study Treatment Start Date $\leq$ AE Start Date $\leq$ Study Treatment Stop Date + 2 days |
| Post-Treatment | If AE onset date is after the treatment stop date + 2 days AE Start Date > Study Treatment Stop Date + 2 days |
| AE Onset Time<br>Since First Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 day Missing otherwise |
| AE Duration<br>(Days) | AE Resolution Date – AE Onset Date + 1 day |
| AE Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

## 10.4 Appendix 4: Data Display Standards & Handling Conventions

#### 10.4.1 Study Treatment & Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Study Part | | Cohort | Data display for reporting |
| | Code | Description | Description <sup>[2]</sup> |
| 1 | 1 | Moderate Hepatic Impairment | Cohort 1 |
| 1 | 2 | Matched Healthy Controls for Moderate Hepatic Impairment | Cohort 2 |
| 2 | 3 | Mild Hepatic Impairment / Severe Hepatic Impairment <sup>[1]</sup> | Cohort 3 |
| 2 | 4 | Matched Healthy Controls for Mild Hepatic Impairment / Matched Healthy Controls for Severe Hepatic Impairment <sup>[1]</sup> | Cohort 4 |

<sup>[1]</sup> Either Mild or Severe Hepatic Impairment participants will be selected based on part 1 results.

#### 10.4.2 Baseline Definition & Derivations

#### 10.4.2.1 Baseline Definitions

For all endpoints (except as noted in Table 9) the baseline value will be the latest non-missing pre-dose assessment. If there are multiple assessments collected on the same scheduled time, the average of these assessments will be used, unless otherwise stated.

Table 10 Baseline Definitions

| Dovomotov | Study Asse | Baseline Used in | | |
|---|---|---|---|---|
| Parameter | Screening | Day -1 | Day 1<br>(Pre-Dose) | Data Display |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | Χ | | Day -1 |
| Haematology | Х | | | Screening |
| Clinical Chemistry | Х | | | Screening |
| Pharmacodynamic | | | | |
| EPO blood sampling | | | Х | Pre-Dose |

<sup>[2]</sup> The word "Cohort" may be omitted from displays in order to limit wrapping

#### 10.4.2.2 Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.2.1 Baseline Definitions will be
  used for derivations for endpoints / parameters and indicated on summaries. Unless otherwise stated, if
  baseline data is missing or post-dose data is missing no derivation will be performed.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.4.3 **Reporting Process & Standards**

#### **Reporting Process** Software The currently supported versions of SAS 9.3 or latest software will be used. Reporting Area HARP Server : UK1SALX00175 HARP Area : arenv/arprod/GSK1278863/mid200231/final QC Spreadsheet : areny/arwork/GSK1278863/mid200231/final/documents **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated only for SAC.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - o Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate (see Section 4.1).

#### **Reporting Standards**

- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - o Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables, unless otherwise stated.
- Unscheduled visits will not be included in figures.

| | All unscheduled visits will be included in listings. |
|---|---|
| Descriptive Summary | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic and Pharmacodynamic Concentration Data | |
| Descriptive Summary<br>Statistics | Refer to IDSL Statistical Principle 6.06.1 and Standards for the Transfer and Reporting of PK and PD Data using HARP. For NQ values, refer to GUI_51487. |
| Reporting of Pharmace | okinetic Parameters |
| Descriptive Summary<br>Statistics.<br>(Log <sub>e</sub> Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log transformed data and %CVb will be reported. CVb (%) = √ (exp(SD²) - 1) * 100 [NOTE: SD = SD of loge transformed data] |
| Parameters Not Being | %AUCex and Tmax |
| Loge Transformed | %AUCex and imax |
| Summary Tables | Cmax, Tmax, AUC(0-t), AUC (0- $\infty$ ), t1/2, and %AUCex as data permit. The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of $\lambda z$ . |
| Summary of Statistical analysis | Geometric mean ratio of hepatic impaired : healthy, point estimate and an associated 90% CI. |
| Listings | Include PK Parameters Cmax, Tmax, AUC(0-t), AUC (0- $\infty$ ), and t1/2 as data permit. Include the first point, last point and number of points used in the determination of $\lambda z$ . |
| Reporting of Pharmac | odynamic Parameters |
| Descriptive Summary Statistics | N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum and maximum |
| Parameters | Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) |
| Summary Tables | Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) as data permit |
| Listings | Include PD Parameters Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) as data permit |
## **Reporting Standards**

## **Graphical Displays**

• Refer to IDSL Statistical Principles 7.01 to 7.13 and Standards for the Transfer and Reporting of PK and PD Data using HARP.

#### 10.5 Appendix 5: Derived and Transformed Data

#### 10.5.1 General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- The worst finding/interpretation associated with multiple measurements as the finding/interpretation for that time point.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from Treatment start date:
  - Ref Date = Missing
- → Day = Missing
- Ref Date < Treatment start Date → Study Day = Ref Date Treatment start Date
- Ref Data ≥ Treatment start Date → Study Day = (Ref Date Treatment start Date) + 1

#### 10.5.2 **Study Population**

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### 10.5.3 Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places = '< x' becomes x 0.01

#### **Laboratory Parameters**

- Example 2: 1 Decimal Places = '> x' becomes x + 0.1
- Example 3: 0 Decimal Places = '< x' becomes x − 1</li>

#### **ECG Parameters**

#### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then :

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^{3} \right] * 1000$$

- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.
- Machine read values of RR should not be replaced with derived values.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **AEs**

#### **AEs OF Special Interest**

- Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis
- Death, MI, stroke, heart failure, thromboembolic events, thrombosis of vascular Access
- Cardiomyopathy
- Pulmonary artery hypertension
- Cancer-related mortality and tumour progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of rheumatoid arthritis

# 10.6 Appendix 6: Premature Withdrawals & Handling of Missing Data

#### 10.6.1 Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A completed subject is one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All subjects who withdraw prematurely from the study will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR).</li> <li>All available data collected up until the point of withdrawal, and the follow-up visits will be used in the analyses and will be listed and all available planned data will be included in the summaries according to the populations defined in Section 4 unless otherwise specified.</li> </ul> |

## 10.6.2 Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank<br/>fields on the collection instrument:</li> </ul> |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.6.2.1 Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | Missing Start Day: First of the month will be used unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered On-treatment as per |

| Element | Reporting Detail |
|---|---|
| | Appendix 3: Treatment States and Phases). |
| | <ul> <li><u>Missing Stop Day</u>: Last day of the month will be used, unless this is after the<br/>stop date of study treatment; in this case the study treatment stop date will<br/>be used.</li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| | <ul> <li>AEs with entirely missing or unknown start dates will be assumed to be on-<br/>treatment for reporting.</li> </ul> |
| | AEs with missing end dates are not anticipated to affect reporting. |

## 10.6.2.2 Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the<br/>full date cannot be ascertained, the following assumptions will be made for<br/>calculating the time to onset and the duration of the event:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month, unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered on-treatment as per Appendix 3: Treatment States).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month, unless this is after the stop date of study treatment; in this case the study</li> </ul> |
| | treatment stop date will be used. |
| | The recorded partial date will be displayed in listings. |

## 10.6.2.3 Handling of PK Concentration Data

| Element | Reporting Detail |
|---|---|
| General | The PK population will be used for the concentration listing, summaries and plotting of the individual concentration-time profiles. |
| | <ul> <li>PK assay results from samples collected from a subject with vomiting occurring within 2 times the median Tmax will not be considered as evaluable.</li> <li>For missing and NQ values, refer to GUI_51487.</li> </ul> |

## 10.6.2.4 Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|------------|--------------------------------------------------|
| Imputation | No imputation will be performed for missing data |

# 10.7 Appendix 7: Values of Potential Clinical Importance

## 10.7.1 Laboratory Values

Laboratory Values of Potential Clinical Importance (Healthy subjects)

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory | Units | Category | Clinical Concern Range | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | >0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | >25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell<br>Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory | Units | Category | Clinical Concern Range | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | > 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

10.7.2 ECG

## ECG Values of Potential Clinical Importance (Healthy subjects)

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

### ECG Values of Potential Clinical Importance (Hepatic Impaired Subjects)

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | > 480 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 |

### 10.7.3 Vital Signs

Vital Sign Values of Potential Clinical Importance (Healthy Subjects)

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate bpm | | < 40 | > 110 |

### CONFIDENTIAL

200231

## Vital Sign Values of Potential Clinical Importance (Hepatic Impaired Subjects)

| Vital Sign Parameter Units | | Clinical Concern Range | |
|-------------------------------|------|------------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 90 | > 160 |
| Diastolic Blood Pressure mmHg | | < 45 | > 95 |
| Heart Rate bpm | | < 50(females) and <45(males) | > 100 |

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

| Endpoint(s) | <ul> <li>PK End points AUC(0-t), AUC (0-∞), Cmax, and t½</li> </ul> |
|---|---|
| Analysis | ANOVA (primary) and ANCOVA (sensitivity) |

#### **Assumptions:**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

# 10.9. Appendix 9: Abbreviations & Trade Marks

### 10.9.1 Abbreviations

| λz | Terminal phase rate constant |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| Ae | Excretion of unchanged drug |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotransferase (SGPT) |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| AUC (0-∞) | Area under the concentration-time curve extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last |
| | time of quantifiable concentration within a subject across all treatments |
| %AUCex | The percentage of AUC $(0-\infty)$ obtained by extrapolation |
| BMI | Body mass index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CKD | Chronic kidney disease |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling and Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CPSSO | Clinical Pharmacology Sciences and Study Operations |
| CRF | Case Report Form |
| $CV_b$ | Coefficient of Variation (Between) |
| DBR | Database Release |
| DP's | Decimal places |
| ECG | Electrocardiogram |
| Emax | Maximum observed effect |
| EPO | Erythropoietin |
| FSH | Follicle stimulating hormone |
| fu | Fraction unbound in plasma |
| GSK | GlaxoSmithKline |
| h | Hour |
| HARP | Harmonized Analysis and Reporting Process |
| Hg | Mercury |
| HI | Hepatic Impairment |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| kg | Kilogram |
| L | Litres |
| mg | Milligram |
| mL | Millilitre |

| mm | Millimetre |
|---|---|
| MM | Mixed Model |
| nm | Nanometer |
| NOAEL | No Observed Adverse Effect Level |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PPD | Pharmaceutical Product Development |
| QSI | Quantitative Sciences India |
| QTc | Electrocardiogram QT interval corrected for heart rate |
| QTcF | Electrocardiogram QT interval corrected for heart rate using Fridericia's |
| | formula |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious adverse event(s) |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |
| SGOT | Serum glutamic-oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SPDS | Statistics, Programming and Data Sciences |
| t½ | Terminal phase half-life |
| Tmax | Time of occurrence of Cmax |
| ULN | Upper Limit of Normal |

## 10.9.2 Trademarks

| Trademarks of the GlaxoSmithKline group of companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.10 Appendix 10: List of Data Displays

## 10.10.1 Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.11 | N/A |
| Safety | 2.1 to 2.19 | N/A |
| Pharmacokinetic | 3.1 to 3.9 | 3.1 to 3.3 |
| Pharmacodynamic | 4.1 to 4.2 | 4.1 to 4.3 |
| Section Listings | | ings |
| ICH Listings | 1 to 47 | |

## 10.10.2 Deliverable

| Delivery | Description |
|----------|-------------------------------------|
| IA | Interim Analysis Complete |
| SAC | Final Statistical Analysis Complete |

# 10.10.3 Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | t Disposition | | | | |
| 1.1 | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| 1.3 | Enrolled | DV1 | Summary of Important Protocol Deviations | | SAC |
| Demog | raphy | | | | |
| 1.4 | Safety | SAFE_T1 | Summary of Child-Pugh Score | | SAC |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.6 | Enrolled | DM11 | Summary of Age Ranges | | SAC |
| 1.7 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.8 | Safety | DM6 | Summary of Race and Racial Combination Details | | SAC |
| 1.9 | Enrolled | SP1A | Summary of Study Population | | SAC |
| 1.10 | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC |
| Medica | I/Surgical Histo | ory & Concomitan | t Medications | · | |
| 1.11 | Safety | CM1 | Summary of Concomitant Medications | | SAC |

## 10.10.4 Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.1 | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.2 | Safety | AE1CP | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.3 | Safety | AE1CP | Summary of Adverse Events Leading to Withdrawal from Study | | SAC |
| 2.4 | Safety | AE1CP | Summary of Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.5 | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.6 | Safety | AE15 | Summary of Common (>=25%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| Labora | tory Measurem | ents | | | |
| 2.7 | Safety | LB1 | Summary of Chemistry Values | | SAC |
| 2.8 | Safety | LB1 | Summary of Chemistry Changes from Baseline | | SAC |
| 2.9 | Safety | LB17 | Summary of Worst Case Chemistry Results Relative to Potential Clinical Importance Criteria Post-Baseline Relative to Baseline | | SAC |
| 2.10 | Safety | LB1 | Summary of Haematology Values | | SAC |
| 2.11 | Safety | LB1 | Summary of Haematology Changes from Baseline | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12 | Safety | LB17 | Summary of Worst Case Haematology Results Relative to Potential Clinical Importance Criteria Post-Baseline Relative to Baseline | | SAC |
| Electro | cardiograms | | | | |
| 2.13 | Safety | EG1 | Summary of ECG Findings | | SAC |
| 2.14 | Safety | EG2 | Summary of ECG Values | | SAC |
| 2.15 | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC |
| 2.16 | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 2.17 | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| Vital Si | gns | | | | · |
| 2.18 | Safety | VS1 | Summary of Vital Signs | | SAC |
| 2.19 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC |

#### 10.10.5 Pharmacokinetic Tables

| Pharma | acokinetic : Tak | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration Tab | le | | | |
| 3.1 | PK | PKCT1 | Summary of Daprodustat and Metabolites Plasma<br>Pharmacokinetic Concentration-Time Data | | SAC |
| 3.2 | PK | PKCT1 | Summary of Daprodustat Unbound Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| PK Der | ived Parameter | rs | | • | |
| 3.3 | PK | PKPT4 | Summary of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters (Non-Transformed) | Parameters with units | SAC |
| 3.4 | PK | PKPT4 | Summary of Derived Daprodustat Unbound Plasma<br>Pharmacokinetic Parameters (Non-Transformed) | Parameters with units | SAC |
| 3.5 | PK | PKPT4 | Summary of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters (Ln-Transformed) | Parameters with units | SAC |
| 3.6 | PK | PKPT4 | Summary of Derived Daprodustat Unbound Plasma Pharmacokinetic Parameters (Ln-Transformed) | Parameters with units | SAC |
| PK Ana | alysis Tables | | | • | |
| 3.7 | PK | PKPT3 | Statistical Analysis of Daprodustat and Metabolites Plasma<br>Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-t), AUC(0-∞), Cmax, t½, free<br>AUC(0-t), free AUC(0-∞) and free<br>Cmax | SAC |
| 3.8 | PK | PKPT3 | Sensitivity Analysis of Daprodustat and Metabolites Plasma<br>Pharmacokinetic Parameters: Analysis of Covariance<br>(ANCOVA) | AUC(0-t), AUC(0-∞), Cmax, t½, free AUC(0-t), free AUC(0-∞) and free Cmax | SAC |
| 3.9 | PK | PK_T1 | Statistical Analysis of Daprodustat and Metabolites Tmax | | SAC |

## 10.10.6 Pharmacokinetic Figures

| Pharmacokinetic : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ual Concentrati | on Plots | | | |
| 3.1 | PK | PKCF1P | Individual Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Paginate by cohort and analyte | SAC |
| Mean / | Median Concer | ntration Plots | | | |
| 3.2 | PK | PKCF2 | Mean Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | SAC |
| 3.3 | PK | PKCF3 | Median Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | SAC |

# 10.10.7 Pharmacodynamic Tables

| Pharmacodynamic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PD Con | centration Dat | a | | | |
| 4.1 | PD | PKCT1 | Summary of Erythropoietin Plasma Pharmacodynamic Concentration-Time Data | | SAC |
| PD Deri | PD Derived Parameter | | | | |
| 4.2 | PD | PKPT4 | Summary of Derived Erythropoietin Plasma Pharmacodynamic Parameters | Parameters with units | SAC |

# 10.10.8 Pharmacodynamic Figures

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Programming Notes | | Deliverable<br>[Priority] |
| Individu | ual Concentrati | on Plots | | | |
| 4.1 | PD | PKCF1P | Individual Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Paginate by cohort | SAC |
| Mean / I | Median Concer | ntration Plots | | | |
| 4.2 | PD | PKCF2 | Mean Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | SAC |
| 4.3 | PD | PKCF3 | Median Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | SAC |

## 10.10.9 ICH Listings

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | • |
| 1 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 2 | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 3 | Enrolled | DV2 | Listing of Important Protocol Deviations | | SAC |
| 4 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Demog | Demography | | | | |
| 5 | Safety | SAFE_L1 | Listing of Child-Pugh Classification and Treatment Assignment | | SAC |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6 | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 7 | Safety | DM9 | Listing of Race | | SAC |
| 8 | Enrolled | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| Medica | I/Surgical Histo | ory & Concomitan | t Medications | , | |
| 9 | Safety | MH2 | Listing of Medical Conditions | | SAC |
| 10 | Safety | CM3 | Listing of Concomitant Medications | | SAC |
| Exposi | ire | I | | | - |
| 11 | Safety | EX3 | Listing of Exposure Data | | SAC |
| Advers | e Events | l | | | 1 |
| 12 | Safety | AE2 | Listing of Relationship between System Organ Class and Verbatim Text | | SAC |
| 13 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 14 | Safety | AE8CP | Listing of All Adverse Events | | SAC |
| 15 | Safety | AE8CP | Listing of Drug-Related Adverse Events | | SAC |
| 16 | Safety | AE8CPA | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | SAC |
| 17 | Safety | AE8CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| 18 | Safety | AE8CP | Listing of Liver Adverse Events | Conditional display | SAC |
| 19 | Safety | AE8CP | Listing of Cardiovascular Adverse Events | Conditional display | SAC |
| 20 | Safety | AE8CP | Listing of Adverse Events of Special Interest | Conditional display | SAC |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory Measurem | ents | | | |
| 21 | Safety | LB13 | Listing of Laboratory Tests and Associated Reference Ranges | | SAC |
| 22 | Safety | LB5 | Listing of Chemistry Values of Potential Clinical Importance | | SAC |
| 23 | Safety | LB5 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 24 | Safety | LB5 | Listing of Haematology Values of Potential Clinical Importance | | SAC |
| 25 | Safety | LB5 | Listing of All Haematology Data for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 26 | Safety | UR2A | Listing of Urinalysis Data | | SAC |
| Electro | cardiograms | l | | | |
| 27 | Safety | EG5 | Listing of Abnormal ECG Findings | | SAC |
| 28 | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC |
| 29 | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC |
| 30 | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| Vital Si | gns | | | | • |
| 31 | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | | SAC |
| 32 | Safety | VS4 | Listing of All Vital Signs for Subjects with Any Value of Potential Clinical Importance | | SAC |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | tion IDSL / TST ID / Example Shell Title | | Programming Notes | Deliverable<br>[Priority] |
| Liver E | vents | | | | |
| 33 | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | Conditional display | SAC |
| 34 | Safety | SU2 | Listing of Alcohol Intake for Subjects with Liver Stopping Events | Conditional display | SAC |
| 35 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional display | SAC |
| 36 | Safety | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | Conditional display | SAC |
| 37 | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional display | SAC |
| 38 | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional display | SAC |
| Pharma | acokinetic | | | | |
| 39 | PK | PKCL1P | Listing of Daprodustat and Metabolites Plasma Pharmacokinetic Concentration-Time Data | Please list all the concentration data including unscheduled | SAC |
| 40 | PK | PKCL1P | Listing of Daprodustat Unbound Plasma Pharmacokinetic Concentration-Time Data | Please list all the concentration data including unscheduled | SAC |
| 41 | PK | PKPL1P | Listing of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | Parameters with units | SAC |
| 42 | PK | PKPL1P | Listing of Derived Daprodustat Unbound Plasma Pharmacokinetic Parameters | Parameters with units | SAC |
| 43 | PK | N/A | RAW SAS Output from Statistical Analysis of Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | | SAC |
| 44 | PK | N/A | RAW SAS Output from Sensitivity Analysis of Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | | SAC |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 45 | PK | N/A | RAW SAS Output from Statistical Analysis of Daprodustat and Metabolites Tmax | | SAC |
| Pharma | codynamic | | | | |
| 46 | PD | PKCL1P | Listing of Erythropoietin Plasma Pharmacodynamic Concentration-Time Data | Please list all the concentration data including unscheduled | SAC |
| 47 | PD | PKPL1P | Listing of Derived Erythropoietin Plasma Pharmacodynamic Parameters | Parameters with units | SAC |

| Division | · | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | ÷ | A Phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with hepatic impairment and matched, healthy control participants with normal hepatic function |
|---|---|---|
| <b>Compound Number</b> | : | GSK1278863 |
| Effective Date | : | 15-SEP-2018 |

#### **Description:**

- The purpose of this reporting and analysis plan (RAP) is to describe the planned analyses and output to be included in Clinical Pharmacology Study Report for Protocol 200231.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.
- This version of the RAP includes amendments to the originally approved RAP (22-Nov-2017)

#### **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Associate Manager Statistics, ([Future Pipeline Discovery, Quantitative Sciences India], Clinical Statistics) | NA | NA |
| Manager ([Clinical Pharmacology, Clinical Pharmacology, QSCi, PCPS, R&D]) | 12-Sep-2018 | e-Signature |
| Pharmacokineticist (Biostatistics, PPD) | 05-Sep-2018 | email |
| Biostatistician (Early Development Services, PPD) | 05-Sep-2018 | email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

#### The GlaxoSmithKline group of companies

### **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Statistics Director (Future Pipeline Discovery, RD PCPS Qsci Clinical Statistics 5D) | 12-Sep-2018 | e-Signature |
| PPD | | |
| Principal Data Manager ([Future Pipeline Discovery, CPSSO Data Management]) | 11-Sep-2018 | e-Signature |
| PPD | | |
| Clinical Development Manager ([Future Pipeline Discovery, RD PCPS CPSSO 1C]) | 11-Sep-2018 | e-Signature |
| PPD | | |
| Senior Director ([Future Pipeline Discovery,<br>Clinical Development, RD MPC HUP]) | 14-Sep-2018 | e-Signature |
| PPD | | |
| Biostatistics and Programming Manager, ([Future Pipeline Discovery, Quantitative Sciences India], Clinical Programming) | 12-Sep-2018 | e-Signature |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Biostatistics and Programming Manager, ([Future Pipeline Discovery, Quantitative Sciences India], Clinical Statistics) | 12-Sep-2018 | e-Signature |
| Programming Manager, ([Future Pipeline Discovery, RD Qsci Clinical Programming Metabolic], Clinical Programming) On behalf of PPD Head QSI, (R&D Projects Clinical Platforms and Sciences, SPDS) | 12-Sep-2018 | e-Signature |

### **TABLE OF CONTENTS**

| | | | | | | PAGE |
|---|---|---|---|---|---|---|
| 1. | | | | | POSIS | |
| | 1.1. | RAP Am | endments | | | 8 |
| 2. | SLIMIN | IARY OF | KEA DBU. | TOCOL INEC | DRMATION | ۵ |
| ۷. | 2.1. | | | | it(s) | |
| | 2.2. | | | | | |
| | 2.3. | | | | | |
| 3. | PLAN | | | | | |
| | 3.1. | | | | | |
| | 3.2. | Final Ana | alyses | | | 12 |
| 4. | | | | | | |
| | 4.1. | Protocol | Deviations | 3 | | 14 |
| 5. | | | | | YSES AND DATA HANDLING | 14 |
| 6. | | | | | | |
| | 6.1. | Overviev | v of Planne | ed Analyses . | | 15 |
| 7. | | _ | | | | |
| | 7.1. | | | | | |
| | 7.2. | 7.2.1. | | | Pharmacokinetic Analyses | |
| | | 1.4.1. | 7.2.1.1. | | entration Measures | |
| | | | 7.2.1.2. | | kinetic Parameters | |
| | | | | 7.2.1.2.1. | | |
| | | | | | Parameters | 17 |
| | | | | 7.2.1.2.2. | | |
| | | | | | Pharmacokinetic Parameters | |
| | 7.3. | | odynamic | Analyses | | <mark>20</mark> |
| | | 7.3.1. | Overview | of Planned I | Pharmacodynamic Analyses | 20 |
| | | | 7.3.1.1. | | dynamic Parameters | 21 |
| | | | | 7.3.1.1.1. | , | |
| | | | | | Parameters | 21 |
| 8. | SAFE | TY ANALY | /SES | | | 22 |
| | 8.1. | | | | vents Analyses | |
| | 8.2. | | | | boratory Analyses | |
| | 8.3. | | | | ety Analyses | |
| 9. | REFE | RENCES. | | | | 25 |
| 10. | APPE | NDICES | | | | 26 |
| | 10.1. | | | | Management | |
| | 10.2. | Appendix | x 2: Time 8 | & Events | - | 28 |
| | | 10.2.1. | Protocol [ | Defined Time | e & Events | <mark>28</mark> |
| | 10.3. | Appendix | x 3: Treatm | nent States | | 30 |


| 2 | n | Λ | 23 | 2 |
|---|---|---|------------|----|
| | U | u | <b>Z</b> . | וכ |

| | 10.3.1. | Treatment | States for AE Data | 30 |
|---|---|---|---|---|
| 10.4. | Appendix | 4: Data Dis | splay Standards & Handling Conventions | 31 |
| | 10.4.1. | | lay Descriptors | |
| | 10.4.2. | | efinition & Derivations | |
| | | | Baseline Definitions | 31 |
| | | 10.4.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | 32 |
| | 10.4.3. | | Process & Standards | |
| 10.5. | | | and Transformed Data | |
| | 10.5.1. | | | |
| | 10.5.2. | | ulation | |
| 40.0 | 10.5.3. | | Maria I and a second se | |
| 10.6. | | | ure Withdrawals & Handling of Missing Data | |
| | 10.6.1. | | Withdrawals | |
| | 10.6.2. | | f Missing Data | |
| | | | Handling of Missing Dates | |
| | | | Handling of Partial Dates | |
| | | | Handling of PK Concentration Data Handling of Missing Data for Statistical | 39 |
| | | | Analysis | 30 |
| 10.7. | Annendiy | 7: Values ( | of Potential Clinical Importance | عد<br>۸۵ |
| 10.7. | 10.7.1. | l ahoratory | Values | 40 |
| | 10.7.1. | • | values | |
| | 10.7.2. | | | |
| 10.8. | | | Checking and Diagnostics for Statistical | |
| 10.0. | | | | 44 |
| 10.9. | | | ations & Trade Marks | |
| | 10.9.1. | | ons | |
| | 10.9.2. | | S | |
| 10.10. | Appendix | | Data Displays | |
| | | | ay Numbering | |
| | | | ) | |
| | 10.10.3. | Study Popu | ulation Tables | 48 |
| | 10.10.4. | Safety Tab | les | 49 |
| | 10.10.5. | Pharmacol | kinetic Tables | 51 |
| | | | kinetic Figures | |
| | | | dynamic Tables | |
| | 10.10.8. | Pharmacoo | dynamic Figures | <u>5</u> 3 |
| | 10.10.9. | ICH Listing | S | 54 |

## 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe: |
| | <ul> <li>The planned analyses and output to be included in the Clinical<br/>Pharmacology Study Report for Protocol 200231. This RAP is intended to<br/>describe the safety and pharmacokinetic (PK) analyses required for the<br/>study which will be provided to the study team members to convey the<br/>content of the reporting efforts, specifically Statistical Analysis Complete<br/>(SAC).</li> </ul> |
| Protocol | This RAP is based on amended protocol (Dated: [15-Nov-2017]) for study 200231 [GlaxoSmithKline Document Number: 2016N305941_01]. |
| Primary<br>Objectives | <ul> <li>To compare plasma PK parameters of daprodustat and its six metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13)) in participants with hepatic impairment to healthy controls matched in gender, age, and body mass index (BMI).</li> <li>To evaluate the impact of hepatic impairment on the plasma protein binding and unbound concentration of daprodustat and its metabolites in plasma</li> </ul> |
| Primary<br>Endpoints | <ul> <li>Daprodustat and its metabolites in plasma area under the concentration-time curve from time zero (predose) extrapolated to infinite time [AUC (0-∞)], percentage of AUC (0-∞) obtained by extrapolation (%AUCex), time zero (predose) to time of last quantifiable concentration [AUC(0-t)], maximum observed concentration (Cmax) following a single oral dose of daprodustat, apparent terminal phase half-life (t½), and time of occurrence of Cmax (Tmax) following a single oral dose of daprodustat.</li> </ul> |
| | Unbound concentration and unbound fraction in plasma of daprodustat and its metabolites at 3, 12 and 24 h post dose (as data permit) |
| Secondary<br>Objectives | To characterize the effect of hepatic impairment on the pharmacodynamics (PD) effect of daprodustat. |
| | To assess the safety and tolerability of a single 6 mg dose of daprodustat. |
| Secondary<br>Endpoints | Maximum observed erythropoietin concentration (Cmax, EPO), Time of the maximum observed erythropoietin concentration (Tmax, EPO) and erythropoietin area under the concentration-time curve from time zero (predose) to the last time of quantifiable erythropoietin concentration [AUC (0-t, EPO)]. |
| | Safety and tolerability parameters, including adverse events and clinical laboratory tests. |

## Overview **Key Elements of the Reporting and Analysis Plan** Study Design A phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with moderate (Part 1) and either mild or severe (Part 2) hepatic impairment and matched, healthy control participants with normal hepatic function. Part 1: Part 1 will include 2 cohorts. Cohort 1 includes participants with moderate hepatic impairment, and Cohort 2 includes matched healthy control participants. Healthy control participants (n=8) will be matched in gender, age (±10 years), and BMI (±15%) to participants with moderate hepatic impairment (n=8; Child-Pugh score of 7-9). All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state. Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 1 of the study. Part 2: Part 2 will include 2 cohorts. Cohort 3 includes participants with either mild or severe hepatic impairment, and Cohort 4 includes matched healthy control participants. Healthy control participants (n=8) will be matched in gender, age (±10 years), and BMI (±15%) to participants with either mild impairment (Child-Pugh score of 5-6) or participants with severe impairment (Child-Pugh score of 10-13) (n=8). All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state. Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 2 of the study. All participants' total involvement with the study will be up to 7 weeks. Planned An informal interim analysis of the primary PK endpoints of AUC $(0-\infty)$ , Analyses AUC(0-t) and Cmax will be conducted for completion of Part 1 of the study. The final planned analyses will be performed, as defined in this RAP document, after database freeze has been declared. Safety and PK/PD data will be presented in tabular and/or graphical format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards.

| Overview | Key Elements of the Reporting and Analysis Plan |
|---|---|
| Analysis<br>Population | <ul> <li>Screened Population: All participants who were screened will be considered<br/>for this population. This population will be used for summarizing screening<br/>status.</li> </ul> |
| | <ul> <li>Enrolled Population: All participants who were successfully screened and<br/>enrolled for the trial and for whom a record exists on the study database.<br/>This population will be used for summarize number of subjects by Country<br/>and Site ID and age ranges.</li> </ul> |
| | Safety Population: All participants who received at least 1 dose of study medication. This will be the primary population for the safety analyses. |
| | PK Population: All participants in the 'Safety Population' for whom a PK sample has been obtained and analyzed will be included in the PK population. This population will be used in the evaluation of PK data. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PK data. |
| | PD Population: All participants in the 'Safety Population' who had at least 1 PD assessment. PD samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PD data. |
| Hypothesis | No formal hypotheses will be tested. |
| Interim<br>Analyses | An informal interim analysis of the primary PK endpoints AUC (0-∞), AUC(0-t and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria: |
| | ➢ If a < 2-fold change in daprodustat exposure (AUC) is observed in<br>participants with moderate hepatic impairment compared to the<br>healthy matched control group, the study may enrol participants with<br>severe hepatic impairment and a healthy, matched control group. |
| | ▶ If a ≥ 2-fold change in daprodustat exposure (AUC) is observed<br>in participants with moderate hepatic impairment compared to the<br>healthy matched control group, the study may enrol participants with<br>mild hepatic impairment and a healthy, matched control group. |

## 1.1. RAP Amendments

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis I | Plan_Study200231_Final_V1 [22-Nov-2017] |
| Reporting and Analysis I | Plan_Study200231_Amendment_Final_V1 [Insert Date] |
| Section 2.1 | <ul> <li>Second primary objective and associate endpoint adds<br/>daprodustat AND its metabolites to plasma protein binding and<br/>unbound concentration in plasma.</li> </ul> |
| | Secondary PD endpoint is revised to say Cmax, EPO instead of Emax; and specifies AUC(0-t, EPO) instead of AUC(last) |
| Section 10.9.1 | Cmax, EPO added |
| Section 7.2.1.2.2 | Added text determining if there is concentration-dependent protein binding. "If data suggest appreciable differences existing in the results obtained based on the observed total and unbound daprodustat PK plasma concentration data, and if deemed appropriate, the bound fraction (1-Fu) at 3 h, 12 h and 24 h will be analysed using paired t-test comparing 12h versus 3h, 24 h versus 3h and 24 h versus 12h". |
| Section 10.4.1 | Updated heading to match with latest updates in TA and TE. Removed Treatment in heading. Study Treatment & Display Descriptors to Study Displays Descriptors. |
| Section 10.7.1 | PCI laboratory values added for hepatic impairment subjects and updated units for Albumin and Creatinine. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Study Objective(s) and Endpoint(s)

| Objectives | | En | dpoints |
|---|---|---|---|
| Primary Objectives | | Primary Endpoints | |
| • | To compare plasma PK parameters of daprodustat and its six metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13)) in participants with hepatic impairment to healthy controls matched in gender, age, and body mass index (BMI). | | Daprodustat and its metabolites plasma area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC $(0-\infty)$ ], percentage of AUC $(0-\infty)$ obtained by extrapolation (%AUCex), time zero (pre-dose) to last time of quantifiable concentration [AUC $(0-t)$ ], maximum observed concentration (Cmax) following a single oral dose of daprodustat, apparent terminal phase half-life ( $t\frac{1}{2}$ ), and time of occurrence of Cmax (Tmax) following a single oral dose of daprodustat. |
| • | To evaluate the impact of hepatic impairment on the plasma protein binding and unbound concentration of daprodustat and its metabolites in plasma. | • | Unbound concentration and unbound fraction in plasma of daprodustat and its metabolites at 3, 12 and 24 h post dose (as data permit). |
| Se | condary Objectives | Se | condary Endpoints |
| • | To characterize the effect of hepatic impairment on the PD effect of daprodustat. | • | Maximum observed erythropoietin concentration (Cmax, EPO), Time of the maximum observed erythropoietin concentration (Tmax, EPO) and erythropoietin area under the concentration-time curve from time zero (pre-dose) to the last time of quantifiable concentration [AUC (0-t, EPO)]. |
| • | To assess the safety and tolerability of a single 6 mg dose of daprodustat. | • | Safety and tolerability parameters, including adverse events and clinical laboratory tests. |

#### 2.2. Study Design

#### **Overview of Study Design and Key Features**

#### **Design Features**

A phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with moderate (Part 1) and either mild or severe (Part 2) hepatic impairment and matched, healthy control participants with normal hepatic function.

#### Part 1:

Part 1 will include 2 cohorts. Cohort 1 includes participants with moderate hepatic impairment, and Cohort 2 includes matched healthy control participants.

Healthy control participants (n=8) will be matched in gender, age  $(\pm 10 \text{ years})$ , and BMI  $(\pm 15\%)$  to participants with moderate hepatic impairment (n=8; Child-Pugh score of 7-9).

All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state.

Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 1 of the study.

#### Part 2:

Part 2 will include 2 cohorts. Cohort 3 includes participants with either mild or severe hepatic impairment, and Cohort 4 includes matched healthy control participants.

Healthy control participants (n=8) will be matched in gender, age ( $\pm 10$  years), and BMI ( $\pm 15\%$ ) to participants with either mild impairment (Child-Pugh score of 5-6) or participants with severe impairment (Child-Pugh score of 10-13) (n=8).

All participants will receive 6 mg of daprodustat as a single oral dose in the fasted state.

Up to 16 participants (8 in each cohort, excluding possible replacements) will be recruited into Part 2 of the study.

All participant's total involvement with the study will be up to 7 weeks.

#### Dosing

#### Part 1

All participants will be administered 6 mg of daprodustat as a single oral dose, with assessments conducted for up to 48 h post dosing (Please refer to Appendix 2)

| Overview of Study Design and Key Features | |
|---|---|
| | Part 2 If conducted, all participants will be administered 6 mg of daprodustat as a single oral dose, with assessments conducted for up to 48 h post dosing. |
| Treatment<br>Assignment | Part 1 consists of up to 16 participants (8 in each cohort, excluding possible replacements). |
| | Part 2 consists of up to 16 participants (8 in each cohort, excluding possible replacements). |
| | All participants will receive the same treatment of a single oral 6 mg dose of daprodustat. |
| Interim Analyses | <ul> <li>An informal interim analysis of the primary PK endpoints AUC (0-∞),<br/>AUC(0-t) and Cmax will be conducted following completion of Part 1 of<br/>the study, with possible progression to Part 2 based on the following<br/>criteria:</li> </ul> |
| | If a < 2-fold change in daprodustat exposure (AUC) is observed<br>in participants with moderate hepatic impairment compared to<br>healthy matched control group, the study may enrol participants<br>with severe hepatic impairment and a healthy, matched control<br>group. |
| | ▶ If a ≥ 2-fold change in daprodustat exposure (AUC) is<br>observed in participants with moderate hepatic impairment<br>compared to healthy matched control group, the study may<br>enrol participants with mild hepatic impairment and a healthy,<br>matched control group. |

## 2.3. Statistical Hypotheses

No formal hypotheses will be tested for this study. An estimation approach will be used to evaluate the effect of hepatic impairment (i.e., moderate and potentially either mild or severe) on the PK of daprodustat. The primary comparisons of interest are the single dose PK parameters, including Cmax and AUC of daprodustat in each hepatic impaired cohort compared to the normal hepatic function cohort.

The point estimates of the geometric least squares (GLS) mean ratio for the PK parameters and associated 90% confidence intervals (CIs) will be provided for cohort comparisons (hepatically impaired: healthy participants). The PK parameters will be log-transformed prior to analysis and cohort comparisons will be expressed as ratios on the original scale. %AUCex and Tmax and will be summarized descriptively.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

An informal interim analysis of the primary endpoints AUC  $(0-\infty)$ , AUC(0-t) and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria:

- If a < 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with severe hepatic impairment and a healthy, matched control group.
- If a ≥ 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with mild hepatic impairment and a healthy, matched control group.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Screened Population | All participants who were screened will be considered for this population. This population will be used for summarizing screening status. | Screen Failure |
| Enrolled Population | All participants who were successfully screened and enrolled for the trial and for whom a record exists on the study database. This population will be used for summarize number of subjects by Country and Site ID and age ranges. | Study Population |
| Safety Population | All participants who received at least one dose of study medication. This will be the primary population for the safety analyses. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK Population | All participants in the 'Safety Population' for whom a PK sample has been obtained and analyzed will be included in the PK population. This population will be used in the evaluation of PK data. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PK data. | • PK |
| PD Population | All participants in the 'Safety Population' who had at least 1 PD assessment. PD samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded from the analyses of PD data. | • PD |

#### NOTES:

• Please refer to Appendix 10 which details the population to be used for each display being generated.
#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarized and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
  - o This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate listing of all inclusion/exclusion criteria deviations will also be provided.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Treatment States |
| 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population displays will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned study population displays, with full details of data displays being presented in Appendix 10: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Disales Ture | Data Displa | ys Generated |
|---|---|---|
| Display Type | Table | Listing |
| Subject Disposition | | |
| Subject Disposition | Y | |
| Reasons for Screening Failures [1] | Υ | Υ |
| Reasons for Withdrawals | | Υ |
| Important Protocol Deviations | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | | Υ |
| Demography | | |
| Demographic Characteristics | Y | Υ |
| Race & Racial Combinations | Y | Υ |
| Study Populations | Y | Υ |
| Summary of Number of Subjects by Country and Site ID | Υ | |
| Summary of Age Ranges | Y | |
| Summary of Child-Pugh score | Y | Υ |
| Medical/Surgical History & Concomitant Medications | | |
| Medical/Surgical History | | Υ |
| Concomitant Medication | Y | Υ |
| Exposure and Treatment Compliance | | |
| Exposure to Study Treatment | | Υ |

<sup>•</sup> Y = Yes display generated.

<sup>[1]</sup> Conditional displays, if data is available table and listing will be generated.

#### 7. PRIMARY STATISTICAL ANALYSES

### 7.1. Interim Analyses

An informal interim analysis of the primary PK endpoints AUC (0-∞), AUC(0-t) and Cmax will be conducted following completion of Part 1 of the study, with possible progression to Part 2 based on the following criteria:

- If a < 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with severe hepatic impairment and a healthy, matched control group.
- If a ≥ 2-fold change in daprodustat exposure (AUC) is observed in participants with moderate hepatic impairment compared to healthy matched control group, the study may enrol participants with mild hepatic impairment and a healthy, matched control group.

## 7.2. Pharmacokinetic Analyses

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by, or under the direct auspices of Clinical Pharmacology Sciences and Study Operations (CPSSO), GlaxoSmithKline.

The merge of PK concentration data and CRF data will be performed by PPD Programming under the direct auspices of Clinical Programming, GlaxoSmithKline.

Derivation of PK parameters will be performed by PPD PK group under the direct auspices of Clinical Pharmacology Modelling and Simulation (CPMS), GlaxoSmithKline.

Statistical analysis of PK data and parameters will be performed by PPD Statistics and Programming under the direct auspices of Clinical Statistics, GlaxoSmithKline.

#### 7.2.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK population, unless otherwise specified.

Table 3 provides an overview of the planned non-compartmental PK analyses of daprodustat and its six metabolites, (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6) and GSK2531401 (M13)) with full details being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Display Type | Untransformed | | | | | | | | | Log- | Transfo | rme | d | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats<br>Analysis | | Summary | | Individual | | Stats<br>Analysis | | Summary | | Individual | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| PK Concentrations | | | | <b>Y</b> [3] | <b>Y</b> [1] [2] | <b>Y</b> [1] | <b>Y</b> [3] | | | | | | | |
| Plasma PK<br>Parameters | <b>Y</b> [4] | | | Υ | | | Υ | <b>Y</b> [4] | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Logarithmic plots will be created on the same display.
- [2] Separate mean and median plots will be generated.
- [3] Unbound PK Concentrations for Daprodustat and its metabolites will be summarized on a separate display.
- [4] Supportive SAS Output from Statistical Analysis.

#### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3. Reporting Process & Standards).

#### 7.2.1.2. Pharmacokinetic Parameters

#### 7.2.1.2.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 10.4.3. Reporting Process & Standards).
- Plasma concentration-time data for daprodustat and its six predominant metabolites will be analysed by non-compartmental methods according to current working practices with WinNonlin 6.4 or higher.
- Non-compartmental analysis will be performed in accordance with GSK PK Guidance document GUI\_51487.
- All calculations of non-compartmental parameters will be based on actual sampling times recorded during the study.
- PK parameters described in Table 4 will be determined from plasma concentration-time data as data permits.

 Table 4
 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid (daprodustat and its six metabolites). |
| AUC(0-∞) | Area under the concentration-time curve extrapolated to infinity calculated as: |
| | AUC(0-∞) = AUC(0-t) + C(t) / lambda_z<br>(daprodustat and its six metabolites) |
| | where C(t) is the last measurable concentration. |
| %AUCex | The percentage of AUC $(0-\infty)$ obtained by extrapolation (%AUCex) will be calculated as: |
| [AUC (0-∞) – AUC(0-t)] / AUC (0-∞) x 10 | |
| | (daprodustat and its six metabolites) |
| Cmax | Maximum observed plasma concentration, determined directly from the concentration-time data. (daprodustat and its six metabolites) |
| Lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the concentration-time curve. (daprodustat and its six metabolites) |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. (daprodustat and its six metabolites) |
| t½ | Apparent terminal phase half-life will be calculated as: |
| | t½ = In2 / Lambda_z |
| | (daprodustat and its six metabolites) |
| fu | Unbound fraction (fu) of daprodustat and its metabolites will be calculated using the total and unbound plasma concentration of daprodustat and its metabolites generated at 3, 12 and 24 h post dose for both normal and hepatic impaired participants using the following formula: |
| | Fu=Cunbound/Ctotal |
| free AUC(0-t) | AUC(0-t) * fu (daprodustat) |

| Parameter | Parameter Description |
|---------------|-----------------------------|
| free AUC(0-∞) | AUC(0-∞) * fu (daprodustat) |
| free Cmax | Cmax * fu (daprodustat) |

#### 7.2.1.2.2. Statistical Analysis of Pharmacokinetic Parameters

For each of the parameters AUC (AUC( $0-\infty$ ), AUC (0-t) and %AUCex)-total and free, t½, Tmax and Cmax-total and free the following summary statistics will be calculated and tabulated by each cohort:

- Untransformed Data: N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum and maximum.
- Loge-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of loge-transformed data and between subject geometric coefficient of variation (%CVb).
- If data suggest appreciable differences existing in the results obtained based on the observed total and unbound daprodustat PK plasma concentration data, and if deemed appropriate, the bound fraction (1-Fu) at 3 h, 12 h and 24 h will be analysed using paired t-test comparing 12h versus 3h, 24 h versus 3h and 24 h versus 12h.

The following PK statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles). Pharmacokinetic analysis and Statistical analyses of the PK parameter data will be the responsibility of PPD.

### **Planned Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

Plasma primary PK endpoints include AUC (0-t), AUC (0-∞). Cmax and t½, as data permit

#### **Model Specification**

 The log-transformed AUC(0-t), AUC (0-∞), Cmax and t½ values for daprodustat and metabolites will be analyzed separately using analysis of variance (ANOVA) as appropriate to the study design, fitting a fixed effect term for cohort. Point estimates and 90% CIs for the differences of interest (hepatically impaired versus healthy participants) will be constructed using the residual variance.

#### **Model Checking & Diagnostics**

• Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios for the hepatically impaired versus healthy participants and 90% CI for the ratios of AUC (0-t), AUC (0-∞). Cmax and t½ for daprodustat and metabolites.

#### **Planned Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

Tmax

#### **Model Specification**

• If data permit, Tmax will be analyzed nonparametrically using the Mann Whitney U test (Wilcoxon rank sum test). The point estimates and 90% CI for the median differences will be derived for hepatic impairment and healthy participants based on Hodges-Lehmann estimation.

### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• The point estimates and 90% confidence intervals for the median differences will be calculated for the cohort difference (hepatically impaired – healthy participants).

#### **Sensitivity Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

• AUC(0-t), AUC(0-∞), Cmax and t1/2

### **Model Specification**

• The log-transformed AUC(0-t), AUC(0-∞), Cmax and t½ values for daprodustat and metabolites will be analyzed separately using analysis of covariance (ANCOVA) as appropriate to the study design, fitting fixed effect terms for cohort, gender, age and BMI. Point estimates and 90% CIs for the differences of interest (hepatically impaired versus healthy participants) will be constructed using the residual variance.

#### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• Statistical analysis by ANCOVA will be presented in tabular format with geometric mean ratios for the difference between participants with hepatically impairment and healthy participants, and 90% CI for the ratios of AUC(0-t), AUC(0-∞), Cmax and t½ for daprodustat and metabolites.

## 7.3. Pharmacodynamic Analyses

#### 7.3.1. Overview of Planned Pharmacodynamic Analyses

The PD analyses will be based on the PD population, unless otherwise specified.

Table 5 provides an overview of the planned PD analyses, with full details being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Pharmacodynamic Analyses

| Display Type | Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Absolute | | | | | | | Change from Baseline | | | | | | |
| | Stats Analysis | | Sur | nmary | nary Individual | | Stats | | Summary | | Individual | | | |
| | | | | | | | Analysis | | | | | | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| PD Concentrations | | | | Υ | <b>Y</b> [1][2] | <b>Y</b> [1] | Υ | | | | | | | |
| PD Parameters | | | | Υ | Υ | | Υ | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Linear and Semi-Logarithmic plots will be created on the same display.
- [2] Separate mean and median plots will be generated.

### 7.3.1.1. Pharmacodynamic Parameters

#### 7.3.1.1.1. Deriving Pharmacodynamic Parameters

- Although erythropoietin (EPO) is an endogenous substance, the plasma concentrations of erythropoietin will not be corrected for baseline endogenous levels Pharmacodynamic analysis will be performed on uncorrected (absolute erythropoietin concentrations) data only.
- Maximum observed erythropoietin concentration (Cmax, EPO), Time of the
  maximum observed erythropoietin concentration (Tmax, EPO) and area under the
  concentration-time curve from time zero (pre-dose) to the last time of quantifiable
  erythropoietin concentration [AUC (0-t, EPO)] will be listed and summarised if
  data is available.
- Pharmacodynamic parameters described in Table 6 will be determined from plasma absolute erythropoietin concentration-time data as data permits.

Table 6 Derived Pharmacodynamic Parameters

| Parameter | Parameter Description |
|---|---|
| Cmax, EPO | Maximum observed EPO concentration |
| Tmax, EPO | Time of the maximum observed EPO concentration |
| AUC (0-t, EPO) | Area under the concentration-time curve from time zero (pre-dose) to the last time of quantifiable erythropoietin concentration |

#### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

### 8.1. Overview of Planned Adverse Events Analyses

Adverse Events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary and summarized by cohort.

Counting of AEs will be based on the number of subjects – not the number of AEs. For example, if a subject experiences the same AE (i.e. same preferred term) more than once, they are counted only once under the count for the preferred term. If a subject experiences more than one AE in a particular system organ class (SOC), they will only be included once in the count for the SOC, but will appear in the count for each appropriate preferred term within the SOC. Therefore, the sum of the numbers of subjects with each preferred term event within a SOC may exceed the total number of subjects with at least one event.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

| Endpoint / Parameter/ Display Type | Absolute | | |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs | Υ | | Υ |
| Serious AEs | Υ | | Υ |
| Drug Related AEs | Υ | | Y |
| AEs leading to withdrawal | Υ | | Y |
| Summary of Common (>=25%) Non-serious Adverse Events by System Organ Class and Preferred Term | Υ | | |
| Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Υ | | |
| Relationship Between System Organ Class and Verbatim Text | | | Y |
| Subject Numbers for Individual Adverse Events | | | Y |
| AEs of special interest [1] | | | Υ |

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Conditional displays, if data is available listing will be generated.

## 8.2. Overview of Planned Clinical Laboratory Analyses

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 8 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| Display Type | Sur | nmary | Individual | Summary | | Individual |
| | Т | F | L | Т | F | L |
| Chemistry | | | | | | |
| Clinical Chemistry | Υ | | Y | Υ | | |
| Clinical Chemistry (Values<br>Outside the PCI Range) | | | Y | | | |
| Haematology | | | | | | |
| Haematology | Υ | | Υ | Υ | | |
| Haematology (Values Outside the PCI Range) | | | Y | | | |
| Urinalysis | | | | | | |
| Urinalysis | | | Υ | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.3. Overview of Planned Other Safety Analyses

Table 9 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays

Table 9 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ | | Abso | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| Display Type | Sur | nmary | Individual | Sum | mary | Individual |
| | Т | F | L | Т | F | L |
| ECG | | | | | | |
| ECG Findings | Υ | | Y | | | |
| ECG Values | Υ | | Υ | Υ | | |
| ECG Values Outside the PCI Range | | | Υ | | | |
| Maximum QTc Values Post-Baseline<br>Relative to Baseline by Category | | | | Υ | | |
| Maximum Increase in QTc Values Post-<br>Baseline Relative to Baseline by<br>Category | | | | Y | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | |
| Vital Signs Measurements Outside the PCI Range | | | Y | | | |

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9. REFERENCES

GlaxoSmithKline Document Number 2016N305941\_00 (Original – 23-MAY-2017): A Phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with hepatic impairment and matched, healthy control participants with normal hepatic function.

GlaxoSmithKline Document Number 2016N305941\_01 (Amended – 15-NOV-2017): A Phase 1, open-label, non-randomized, parallel group, single-dose adaptive study in adults with hepatic impairment and matched, healthy control participants with normal hepatic function.

GUI\_137354, Information for Authors: Reporting and Analysis Plan (RAP), Global. 2018

GUI\_51487, Non-Compartmental Analysis of Pharmacokinetic Data, CPMS Global. Date: 21-AUG-2018.

SOP\_54838, Development, Review & Approval of Reporting & Analysis Plan (RAP), Global. Date: 22-Aug-2018.

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4: | Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5: | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Treatment States |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General |
| | Study Population |
| | Safety |
| | Pharmacokinetic |
| | Pharmacodynamic |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| | <ul> <li>Handling of Missing Dates</li> </ul> |
| | <ul> <li>Handling of Partial Dates</li> </ul> |
| Section 10.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.9 | Appendix 9 Abbreviations & Trade Marks |
| Section 10.10 | Appendix 10: List of Data Displays |

## 10.1. Appendix 1: Protocol Deviation Management

There are no pre-defined categories leading to exclusion from the PK population but all protocol deviations will be reviewed on a case-by-case basis.

No subjects will be excluded from the safety population.

## 10.2. Appendix 2: Time & Events

## 10.2.1. Protocol Defined Time & Events

| Procedure | Screening <sup>1</sup> | Day -1 | Pre-Dose | 0 h | 0.5 h | t<br>t | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 36 h | 48 h | Follow-up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | Х | | | | | | | | | | | | | | | | | |
| Inclusion & Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | | | | |
| Full physical exam | Х | | | | | | | | | | | | | | | | | |
| Medical<br>history | Χ | | | | | | | | | | | | | | | | | |
| Past/current medications | Х | | | | | | | | | | | | | | | | | |
| Laboratory assessments <sup>3</sup> | Χ | | | | | | | | | | | | | | | | Х | Х |
| Drug/Alcohol<br>Screen | Х | Х | | | | | | | | | | | | | | | | |
| 12-lead ECG | Χ | Χ | | | | | | | | | | | | | | | Χ | Χ |
| Vital Signs and Weight | Х | Х | | | | | | | | | | | | | | | Χ | Х |
| Pregnancy<br>Test | X <sup>4</sup> | X <sup>4</sup> | | | | | | | | | | | | | | | | |
| Females only:<br>Estrogen and<br>FSH <sup>5</sup> | Х | | | | | | | | | | | | | | | | | |

| Procedure | Screening <sup>1</sup> | Day -1 | Pre-Dose | 0 h | 0.5 h | 1 h | 1.5 h | 2 h | 3 h | 4 h | 6 h | 8 h | 10 h | 12 h | 24 h | 36 h | 48 h | Follow-up <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Admission to Unit | | Х | | | | | | | | | | | | | | | | |
| Brief Physical<br>Exam | | Х | | | | | | | | | | | | | | | Х | Х |
| Administration of daprodustat | | | | Х | | | | | | | | | | | | | | |
| PK blood sampling | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Protein binding sample | | | Х | | | | | | Х | | | | | Х | Χ | | | |
| EPO blood sampling | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Adverse<br>Events<br>Assessment | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Χ | Χ | Χ | х |
| Review<br>Concomitant<br>Medications | | Х | х | | | | | | | | | | | | X | | Χ | Х |
| Discharge<br>from Unit | | | | | | | | | | | | | | | | | Х | |

<sup>&</sup>lt;sup>1</sup> All participants will undergo screening assessments within 28 days of enrolment.

<sup>&</sup>lt;sup>2</sup> A follow-up visit will occur 10-14 days after the dose of study treatment.

<sup>&</sup>lt;sup>3</sup> Laboratory assessment guidance can be found in Protocol Appendix 3.

<sup>&</sup>lt;sup>4</sup> For women of childbearing potential that are not using an approved method of contraception (see Protocol Appendix 6), one negative pregnancy test between Day -7 and Day -4 AND another negative pregnancy test on Day -1 is required. Additional guidance can be found in Protocol Section 9.5.5.

<sup>&</sup>lt;sup>5</sup> All females are to have estrogen and FSH measured at screening.

## 10.3. Appendix 3: Treatment States

#### 10.3.1. Treatment States for AE Data

Assessments and events will be classified according to date of occurrence relative to the start and/or stop date of the study treatment.

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before the treatment stop date 2 days |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 2 days |
| Post-Treatment | If AE onset date is after the treatment stop date + 2 days AE Start Date > Study Treatment Stop Date + 2 days |
| AE Onset Time<br>Since First Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 day Missing otherwise |
| AE Duration (Days) | AE Resolution Date – AE Onset Date + 1 day |
| AE Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

• If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

### 10.4.1. Study Display Descriptors

| Study Display Descriptions | | | |
|---|---|---|---|
| Study Part | | Cohort | Data display for reporting |
| | Code | Description | Description [2] |
| 1 | 1 | Moderate Hepatic Impairment | Cohort 1 |
| 1 | 2 | Matched Healthy Controls for Moderate Hepatic Impairment | Cohort 2 |
| 2 | 3 | Mild Hepatic Impairment / Severe Hepatic Impairment <sup>[1]</sup> | Cohort 3 |
| 2 | 4 | Matched Healthy Controls for Mild Hepatic Impairment / Matched Healthy Controls for Severe Hepatic Impairment <sup>[1]</sup> | Cohort 4 |

<sup>[1]</sup> Either Mild or Severe Hepatic Impairment participants will be selected based on part 1 results.

#### 10.4.2. Baseline Definition & Derivations

#### 10.4.2.1. Baseline Definitions

For all endpoints (except as noted in Table 9) the baseline value will be the latest non-missing pre-dose assessment. If there are multiple assessments collected on the same scheduled time, the average of these assessments will be used, unless otherwise stated.

Table 10 Baseline Definitions

| Devenuetor | Study Asse | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| Parameter | Screening Day -1 Day 1 (Pre-Dose) | | | |
| Safety | | | | |
| 12 Lead ECG & Vital Signs | Х | Х | | Day -1 |
| Haematology | Х | | | Screening |
| Clinical Chemistry | X | | | Screening |
| Pharmacodynamic | | | | |
| EPO blood sampling | | | Х | Pre-Dose |

<sup>[2]</sup> The word "Cohort" may be omitted from displays in order to limit wrapping

#### 10.4.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.4.2.1 Baseline Definitions will be
  used for derivations for endpoints / parameters and indicated on summaries. Unless otherwise stated, if
  baseline data is missing or post-dose data is missing no derivation will be performed.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.4.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | |
| <ul> <li>The currently supported versions of SAS 9.3 or latest software will be used.</li> </ul> | |
| Reporting Area | Reporting Area |
| HARP Server | : UK1SALX00175 |
| HARP Area | : arenv/arprod/GSK1278863/mid200231/final |
| QC Spreadsheet : arenv/arwork/GSK1278863/mid200231/final/documents | |
| Analysis Detecto | Analysis Detects |

#### **Analysis Datasets**

Reporting Process

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated only for SAC.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.

#### **Reporting Standards**

- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate (see Section 4.1).
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables, unless otherwise stated.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| <b>Descriptive Summary S</b> | Statistics |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharmacokinetic and Pharmacodynamic Concentration Data | |
| Descriptive Summary<br>Statistics | Refer to IDSL Statistical Principle 6.06.1 and Standards for the Transfer and Reporting of PK and PD Data using HARP. For NQ values, refer to GUI_51487. |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive Summary<br>Statistics.<br>(Log <sub>e</sub> Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log transformed data and %CVb will be reported. CVb (%) = $\sqrt{(\exp(SD^2) - 1) * 100}$ [NOTE: SD = SD of loge transformed data] |
| Parameters Not Being Loge Transformed | %AUCex and Tmax |
| Summary Tables | Cmax, Tmax, AUC(0-t), AUC (0- $\infty$ ), t1/2, and %AUCex as data permit. The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of $\lambda$ z. |
| Summary of Statistical analysis | Geometric mean ratio of hepatic impaired : healthy, point estimate and an associated 90% CI. |

| Reporting Standards | |
|---|---|
| Listings | Include PK Parameters Cmax, Tmax, AUC(0-t), AUC (0- $\infty$ ), and t1/2 as data permit. Include the first point, last point and number of points used in the determination of $\lambda z$ . |
| Reporting of Pharmacodynamic Parameters | |
| Descriptive Summary Statistics | N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum and maximum |
| Parameters | Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) |
| Summary Tables | Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) as data permit |
| Listings | Include PD Parameters Cmax, EPO, Tmax, EPO and AUC (0-t, EPO) as data permit |
| Graphical Displays | |
| <ul> <li>Refer to IDSL Statistical Principles 7.01 to 7.13 and Standards for the Transfer and Reporting<br/>of PK and PD Data using HARP.</li> </ul> | |

#### 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- The worst finding/interpretation associated with multiple measurements as the finding/interpretation for that time point.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from Treatment start date:
  - Ref Date = Missing
- → Day = Missing
- Ref Date < Treatment start Date → Study Day = Ref Date Treatment start Date
- Ref Data ≥ Treatment start Date → Study Day = (Ref Date Treatment start Date) + 1

#### 10.5.2. **Study Population**

### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### 10.5.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of decimal places in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places = '< x' becomes x 0.01
  - Example 2: 1 Decimal Places = '> x' becomes x + 0.1

### **Laboratory Parameters**

• Example 3: 0 Decimal Places = '< x' becomes x − 1

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.
- Machine read values of RR should not be replaced with derived values.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **AEs**

## **AEs OF Special Interest**

- Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis
- Death, MI, stroke, heart failure, thromboembolic events, thrombosis of vascular Access
- Cardiomyopathy
- Pulmonary artery hypertension
- Cancer-related mortality and tumour progression and recurrence
- Esophageal and gastric erosions
- Proliferative retinopathy, macular edema, choroidal neovascularization
- Exacerbation of rheumatoid arthritis

# 10.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

### 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A completed subject is one who has completed all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All subjects who withdraw prematurely from the study will be documented and the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR).</li> <li>All available data collected up until the point of withdrawal, and the follow-up visits will be used in the analyses and will be listed and all available planned data will be included in the summaries according to the populations defined in Section 4 unless otherwise specified.</li> </ul> |

## 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 10.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | Missing Start Day: First of the month will be used unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered On-treatment as per |

| Element | Reporting Detail |
|---|---|
| | Appendix 3: Treatment States). |
| | <ul> <li><u>Missing Stop Day</u>: Last day of the month will be used, unless this is after the<br/>stop date of study treatment; in this case the study treatment stop date will<br/>be used.</li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| | AEs with entirely missing or unknown start dates will be assumed to be ontreatment for reporting. |
| | AEs with missing end dates are not anticipated to affect reporting. |

## 10.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the<br/>full date cannot be ascertained, the following assumptions will be made for<br/>calculating the time to onset and the duration of the event:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month, unless this is before the start date of investigational<br/>product; in this case the study treatment start date will be used (and hence<br/>the event is considered on-treatment as per Appendix 3: Treatment States).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month,<br/>unless this is after the stop date of study treatment; in this case the study<br/>treatment stop date will be used.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

## 10.6.2.3. Handling of PK Concentration Data

| Element | Reporting Detail |
|---|---|
| General | The PK population will be used for the concentration listing, summaries and plotting of the individual concentration-time profiles. |
| | <ul> <li>PK assay results from samples collected from a subject with vomiting occurring within 2 times the median Tmax will not be considered as evaluable.</li> <li>For missing and NQ values, refer to GUI_51487.</li> </ul> |

## 10.6.2.4. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|------------|--------------------------------------------------|
| Imputation | No imputation will be performed for missing data |

## 10.7. Appendix 7: Values of Potential Clinical Importance

## 10.7.1. Laboratory Values

Laboratory Values of Potential Clinical Importance (Healthy subjects)

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory | Units Category | | Clinical Concern Range | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | >0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| _ | | $\Delta$ from BL | >25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell<br>Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory | Units | Category | Clinical Concern Range | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | > 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## Laboratory Values of Potential Clinical Importance (Hepatic Impaired Subjects)

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory | Units | Category | Clinical Concern Range | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | >0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | >25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell<br>Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Units Category Clinical Concern Range | | | | |
| Parameter | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | > 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 3x ULN |
| AST/SGOT | U/L | High | ≥ 3x ULN |
| AlkPhos | U/L | High | ≥ 3x ULN |
| T Bilirubin | µmol/L | High | ≥ 2xULN |
| | µmol/L | | 2xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 3x ULN ALT |

10.7.2. ECG

## ECG Values of Potential Clinical Importance (Healthy subjects)

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | Change from Baseline | | |
| Increase from Baseline QTc | msec | | > 60 |

## ECG Values of Potential Clinical Importance (Hepatic Impaired Subjects)

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 480 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | Change from Baseline | | |
| Increase from Baseline<br>QTc | msec | | > 60 |

## 10.7.3. Vital Signs

Vital Sign Values of Potential Clinical Importance (Healthy Subjects)

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

## CONFIDENTIAL

200231

## Vital Sign Values of Potential Clinical Importance (Hepatic Impaired Subjects)

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 90 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 95 |
| Heart Rate | bpm | < 50(females) and <45(males) | > 100 |

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

| Endpoint(s) | <ul> <li>PK End points AUC(0-t), AUC (0-∞), Cmax, and t½</li> </ul> |
|---|---|
| Analysis | ANOVA (primary) and ANCOVA (sensitivity) |

#### **Assumptions:**

- For the Mixed Model, model assumptions will be checked, and appropriate adjustments may be applied based on the data.
- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.
- Non-parametric analyses will be conducted if the normality assumption does not hold.

## 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| λz | Terminal phase rate constant |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| Ae | Excretion of unchanged drug |
| AIC | Akaike's Information Criteria |
| ALT | Alanine aminotransferase (SGPT) |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate aminotransferase (SGOT) |
| AUC | Area under concentration-time curve |
| AUC (0-∞) | Area under the concentration-time curve extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time zero (pre-dose) to last |
| | time of quantifiable concentration within a subject across all treatments |
| AUC0-t, | Area under the EPO concentration-time curve from time zero (pre-dose) |
| EPO | to last time of quantifiable EPO concentration within a subject across all |
| | treatments |
| %AUCex | The percentage of AUC $(0-\infty)$ obtained by extrapolation |
| BMI | Body mass index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | |
| CKD | Chronic kidney disease |
| Cmax | Maximum observed concentration |
| Cmax, EPO | Maximum observed EPO concentration |
| CPMS | Clinical Pharmacology Modelling and Simulation |
| CPSR | Clinical Pharmacology Study Report |
| CPSSO | Clinical Pharmacology Sciences and Study Operations |
| CRF | Case Report Form |
| CV <sub>b</sub> | Coefficient of Variation (Between) |
| DBR | Database Release |
| DP's | Decimal places |
| ECG | Electrocardiogram |
| Emax | Maximum observed effect |
| EPO | Erythropoietin |
| FSH | Follicle stimulating hormone |
| fu | Fraction unbound in plasma |
| GSK | GlaxoSmithKline |
| h | Hour |
| HARP | Harmonized Analysis and Reporting Process |
| Hg | Mercury |
| HI | Hepatic Impairment |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |

| kg | Kilogram |
|---|---|
| L | Litres |
| mg | Milligram |
| mL | Millilitre |
| mm | Millimetre |
| MM | Mixed Model |
| nm | Nanometer |
| NOAEL | No Observed Adverse Effect Level |
| PD | Pharmacodynamic |
| PK | Pharmacokinetic |
| PPD | Pharmaceutical Product Development |
| QSI | Quantitative Sciences India |
| QTc | Electrocardiogram QT interval corrected for heart rate |
| QTcF | Electrocardiogram QT interval corrected for heart rate using Fridericia's |
| | formula |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious adverse event(s) |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |
| SGOT | Serum glutamic-oxaloacetic transaminase |
| SGPT | Serum glutamic pyruvic transaminase |
| SPDS | Statistics, Programming and Data Sciences |
| t½ | Terminal phase half-life |
| Tmax | Time of occurrence of Cmax |
| Tmax, EPO | Time of occurrence of Cmax, EPO |
| ULN | Upper Limit of Normal |

## 10.9.2. Trademarks

| | Trademarks of the GlaxoSmithKline group of companies |
|---|------------------------------------------------------|
| Ī | NONE |

| Trademarks not owned by the GlaxoSmithKline group of companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

## 10.10. Appendix 10: List of Data Displays

## 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.11 | N/A |
| Safety | 2.1 to 2.19 | N/A |
| Pharmacokinetic | 3.1 to 3.10 | 3.1 to 3.3 |
| Pharmacodynamic | 4.1 to 4.2 | 4.1 to 4.3 |
| Section | List | ings |
| ICH Listings | 1 to 47 | |

## 10.10.2. Deliverable

| Delivery | Description |
|----------|-------------------------------------|
| DR | Dry Run Complete |
| SAC | Final Statistical Analysis Complete |

## 10.10.3. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1 | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | DR, SAC |
| 1.2 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | DR, SAC |
| 1.3 | Enrolled | DV1 | Summary of Important Protocol Deviations | | DR, SAC |
| Demog | raphy | | | | |
| 1.4 | Safety | SAFE_T1 | Summary of Child-Pugh Score | | DR, SAC |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | DR, SAC |
| 1.6 | Enrolled | DM11 | Summary of Age Ranges | | DR, SAC |
| 1.7 | Safety | DM5 | Summary of Race and Racial Combinations | | DR, SAC |
| 1.8 | Safety | DM6 | Summary of Race and Racial Combination Details | | DR, SAC |
| 1.9 | Enrolled | SP1A | Summary of Study Population | | DR, SAC |
| 1.10 | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | DR, SAC |
| Medica | Medical/Surgical History & Concomitant Medications | | | | |
| 1.11 | Safety | CM1 | Summary of Concomitant Medications | | DR, SAC |

## 10.10.4. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 2.1 | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | | DR, SAC |
| 2.2 | Safety | AE1CP | Summary of Drug-Related Adverse Events by System Organ Class and Preferred Term | | DR, SAC |
| 2.3 | Safety | AE1CP | Summary of Adverse Events Leading to Withdrawal from Study | | DR, SAC |
| 2.4 | Safety | AE1CP | Summary of Serious Adverse Events by System Organ Class and Preferred Term | | DR, SAC |
| 2.5 | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | DR, SAC |
| 2.6 | Safety | AE15 | Summary of Common (>=25%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | DR, SAC |
| Labora | tory Measurem | ents | | 1 | , |
| 2.7 | Safety | LB1 | Summary of Chemistry Values | | DR, SAC |
| 2.8 | Safety | LB1 | Summary of Chemistry Changes from Baseline | | DR, SAC |
| 2.9 | Safety | LB17 | Summary of Worst Case Chemistry Results Relative to Potential Clinical Importance Criteria Post-Baseline Relative to Baseline | | DR, SAC |
| 2.10 | Safety | LB1 | Summary of Haematology Values | | DR, SAC |
| 2.11 | Safety | LB1 | Summary of Haematology Changes from Baseline | | DR, SAC |
| 2.12 | Safety | LB17 | Summary of Worst Case Haematology Results Relative to Potential Clinical Importance Criteria Post-Baseline Relative to Baseline | | DR, SAC |

| Safety : | Safety : Tables | | | |
|---|---|---|---|---|
| Electro | cardiograms | | | |
| 2.13 | Safety | EG1 | Summary of ECG Findings | DR, SAC |
| 2.14 | Safety | EG2 | Summary of ECG Values | DR, SAC |
| 2.15 | Safety | EG2 | Summary of Change from Baseline in ECG Values | DR, SAC |
| 2.16 | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | DR, SAC |
| 2.17 | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | DR, SAC |
| Vital Signs | | | | |
| 2.18 | Safety | VS1 | Summary of Vital Signs | DR, SAC |
| 2.19 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | DR, SAC |

### 10.10.5. Pharmacokinetic Tables

| Pharma | acokinetic : Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | ncentration Tab | le | | | |
| 3.1 | PK | PKCT1 | Summary of Daprodustat and Metabolites Plasma Pharmacokinetic Concentration-Time Data | | DR, SAC |
| 3.2 | PK | PKCT1 | Summary of Daprodustat and Metabolites Unbound Plasma<br>Pharmacokinetic Concentration-Time Data | | DR, SAC |
| PK Der | ived Parameter | S | | | |
| 3.3 | PK | PKPT4 | Summary of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters (Non-Transformed) | Parameters with units | DR, SAC |
| 3.4 | PK | PKPT4 | Summary of Derived Daprodustat Unbound Plasma<br>Pharmacokinetic Parameters (Non-Transformed) | Parameters with units | DR, SAC |
| 3.5 | PK | PKPT4 | Summary of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters (Ln-Transformed) | Parameters with units | DR, SAC |
| 3.6 | PK | PKPT4 | Summary of Derived Daprodustat Unbound Plasma<br>Pharmacokinetic Parameters (Ln-Transformed) | Parameters with units | DR, SAC |
| PK Ana | alysis Tables | | | | |
| 3.7 | PK | PKPT3 | Statistical Analysis of Daprodustat and Metabolites Plasma<br>Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-t), AUC(0-∞), Cmax, t½, free<br>AUC(0-t), free AUC(0-∞) and free Cmax | DR, SAC |
| 3.8 | PK | PKPT3 | Sensitivity Analysis of Daprodustat and Metabolites Plasma<br>Pharmacokinetic Parameters: Analysis of Covariance (ANCOVA) | AUC(0-t), AUC(0-∞), Cmax, t½, free AUC(0-t), free AUC(0-∞) and free Cmax | DR, SAC |
| 3.9 | PK | PK_T1 | Statistical Analysis of Daprodustat and Metabolites Tmax | | DR, SAC |
| 3.10 | PK | PKPT3 | Statistical Analysis of Daprodustat Bound Fraction (1-Fu) in Plasma | | SAC |

## 10.10.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ual Concentrati | on Plots | | | |
| 3.1 | PK | PKCF1P | Individual Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Paginate by cohort and analyte | DR, SAC |
| Mean / I | Median Conce | ntration Plots | | | |
| 3.2 | PK | PKCF2 | Mean Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | DR, SAC |
| 3.3 | PK | PKCF3 | Median Daprodustat and Metabolites Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | DR, SAC |

## 10.10.7. Pharmacodynamic Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PD Con | PD Concentration Data | | | | |
| 4.1 | PD | PKCT1 | Summary of Erythropoietin Plasma Pharmacodynamic Concentration-Time Data | | DR, SAC |
| PD Deri | PD Derived Parameter | | | | |
| 4.2 | PD | PKPT4 | Summary of Derived Erythropoietin Plasma Pharmacodynamic Parameters | Parameters with units | DR, SAC |

## 10.10.8. Pharmacodynamic Figures

| Pharma | Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ual Concentrati | on Plots | | | |
| 4.1 | PD | PKCF1P | Individual Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Paginate by cohort | DR, SAC |
| Mean / I | Median Concer | ntration Plots | | | |
| 4.2 | PD | PKCF2 | Mean Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | DR, SAC |
| 4.3 | PD | PKCF3 | Median Erythropoietin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | All cohorts on one page | DR, SAC |

## 10.10.9. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | <u> </u> |
| 1 | Safety | ES2 | Listing of Reasons for Study Withdrawal | | DR, SAC |
| 2 | Screened | ES7 | Listing of Reasons for Screen Failure | | DR, SAC |
| 3 | Enrolled | DV2 | Listing of Important Protocol Deviations | | DR, SAC |
| 4 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | DR, SAC |
| Demog | raphy | | | | <u> </u> |
| 5 | Safety | SAFE_L1 | Listing of Child-Pugh Classification and Treatment Assignment | | DR, SAC |
| 6 | Safety | DM2 | Listing of Demographic Characteristics | | DR, SAC |
| 7 | Safety | DM9 | Listing of Race | | DR, SAC |
| 8 | Enrolled | SP3 | Listing of Subjects Excluded from Any Population | | DR, SAC |
| Medica | al/Surgical Histo | ory & Concomitan | t Medications | | <u> </u> |
| 9 | Safety | MH2 | Listing of Medical Conditions | | DR, SAC |
| 10 | Safety | CM3 | Listing of Concomitant Medications | | DR, SAC |
| Exposi | ure | 1 | · | • | |
| 11 | Safety | EX3 | Listing of Exposure Data | | DR, SAC |
| Advers | se Events | | | | , |
| 12 | Safety | AE2 | Listing of Relationship between System Organ Class and Verbatim Text | | DR, SAC |

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 13 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | DR, SAC |
| 14 | Safety | AE8CP | Listing of All Adverse Events | | DR, SAC |
| 15 | Safety | AE8CP | Listing of Drug-Related Adverse Events | | DR, SAC |
| 16 | Safety | AE8CPA | Listing of Serious Adverse Events (Fatal & Non-Fatal) | | DR, SAC |
| 17 | Safety | AE8CP | Listing of Adverse Events Leading to Withdrawal from Study | | DR, SAC |
| 18 | Safety | AE8CP | Listing of Liver Adverse Events | Conditional display | DR, SAC |
| 19 | Safety | AE8CP | Listing of Cardiovascular Adverse Events | Conditional display | DR, SAC |
| 20 | Safety | AE8CP | Listing of Adverse Events of Special Interest | Conditional display | DR, SAC |
| Labora | tory Measurem | ents | | | |
| 21 | Safety | LB13 | Listing of Laboratory Tests and Associated Reference Ranges | | DR, SAC |
| 22 | Safety | LB5 | Listing of Chemistry Values of Potential Clinical Importance | | DR, SAC |
| 23 | Safety | LB5 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance | | DR, SAC |
| 24 | Safety | LB5 | Listing of Haematology Values of Potential Clinical Importance | | DR, SAC |
| 25 | Safety | LB5 | Listing of All Haematology Data for Subjects with Any Value of Potential Clinical Importance | | DR, SAC |
| 26 | Safety | UR2A | Listing of Urinalysis Data | | DR, SAC |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Electro | cardiograms | | | | <u> </u> |
| 27 | Safety | EG5 | Listing of Abnormal ECG Findings | | DR, SAC |
| 28 | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | DR, SAC |
| 29 | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | | DR, SAC |
| 30 | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | DR, SAC |
| Vital Si | gns | | | | |
| 31 | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | | DR, SAC |
| 32 | Safety | VS4 | Listing of All Vital Signs for Subjects with Any Value of Potential Clinical Importance | | DR, SAC |
| Liver E | vents | | | | <u> </u> |
| 33 | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping<br>Events | Conditional display | DR, SAC |
| 34 | Safety | SU2 | Listing of Alcohol Intake for Subjects with Liver Stopping Events | Conditional display | DR, SAC |
| 35 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional display | DR, SAC |
| 36 | Safety | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | Conditional display | DR, SAC |
| 37 | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional display | DR, SAC |
| 38 | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional display | DR, SAC |

| ICH : Li | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | acokinetic | | | | |
| 39 | PK | PKCL1P | Listing of Daprodustat and Metabolites Plasma Pharmacokinetic Concentration-Time Data | Please list all the concentration data including unscheduled | DR, SAC |
| 40 | PK | PKCL1P | Listing of Daprodustat and Metabolites Unbound Plasma Pharmacokinetic Concentration-Time Data | Please list all the concentration data including unscheduled | DR, SAC |
| 41 | PK | PKPL1P | Listing of Derived Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | Parameters with units | DR, SAC |
| 42 | PK | PKPL1P | Listing of Derived Daprodustat Unbound Plasma Pharmacokinetic Parameters | Parameters with units | DR, SAC |
| 43 | PK | N/A | RAW SAS Output from Statistical Analysis of Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | | DR, SAC |
| 44 | PK | N/A | RAW SAS Output from Sensitivity Analysis of Daprodustat and Metabolites Plasma Pharmacokinetic Parameters | | DR, SAC |
| 45 | PK | N/A | RAW SAS Output from Statistical Analysis of Daprodustat and Metabolites Tmax | | DR, SAC |
| Pharma | acodynamic | | | | |
| 46 | PD | PKCL1P | Listing of Erythropoietin Plasma Pharmacodynamic Concentration-Time Data | Please list all the concentration data including unscheduled | DR, SAC |
| 47 | PD | PKPL1P | Listing of Derived Erythropoietin Plasma Pharmacodynamic Parameters | Parameters with units | DR, SAC |